Official Title: A Phase 2 Study Evaluating the Efficacy and Safety of VIR-3434 and/or VIR-2218 Containing Regimens in HBeAg-negative Participants with Low Viral Burden of Chronic Hepatitis B Infection (THRIVE)

NCT Number: NCT05612581

Document Date: 26 January 2024, Version 1.0



# PREVAIL PLATFORM CLINICAL STUDY SUB-PROTOCOL B (THRIVE) PROTOCOL AMENDMENT 3

This sub-protocol should be read and conducted in conjunction with the PREVAIL Master Protocol

| Study Title | A Phase 2 Study Evaluating the Efficacy and Safety of VIR-3434 and/or VIR-2218 Containing Regimens in HBeAg-negative Participants with Low Viral Burden of Chronic Hepatitis B Infection (THRIVE) |
|---|---|
| Brief Title | A Phase 2 Study to Evaluate VIR-3434 and/or VIR-2218 Containing Regimens for Treatment of Chronic Hepatitis B Infection |
| Master Study Number | VIR-MHB1-V200 |
| Sub-Study Number | VIR-SHB1-V202 |
| Compounds | VIR-3434 (tobevibart), VIR-2218 (elebsiran), and tenofovir disoproxil fumarate (TDF) |
| Indication | Chronic Hepatitis B Infection |
| Study Phase 2 | |
| Study Sponsor | Vir Biotechnology, Inc.<br>1800 Owens Street, Suite 900<br>San Francisco, CA 94158, USA |
| Regulatory Agency<br>Identifying Numbers | IND: TBD EudraCT: 2022-002014-16 (under Master Protocol) NCT: 05612581 (under Master Protocol) |
| <b>Protocol Date</b> | 26 January 2024, Version 1.0 |

This study will be conducted in compliance with International Council for Harmonisation (ICH) Good Clinical Practice (GCP), including the archiving of essential documents

#### CONFIDENTIALITY STATEMENT

This document contains confidential information that is the property of Vir Biotechnology, Inc. This confidential information is being provided to you, your staff, the applicable Institutional Review Board/Independent Ethics Committee, and applicable regulatory authorities solely for the purpose of evaluating or conducting this clinical study. This confidential information will be protected by you and your staff against disclosure to or use by third parties, except as necessary for the evaluation or conduct of the study.

# **INVESTIGATOR SIGNATURE PAGE**

# VIR BIOTECHNOLOGY, INC 1800 OWENS STREET, SUITE 900 SAN FRANCISCO, CA 94158

#### STUDY ACKNOWLEDGMENT

A Phase 2 Study Evaluating the Efficacy and Safety of VIR-3434 and/or VIR-2218 Containing Regimens in HBeAg-negative Participants with Low Viral Burden of Chronic Hepatitis B Infection (THRIVE)

This sub-protocol has been approved by Vir Biotechnology, Inc. The following signature documents this approval.

| Printed Name | Signature and Date |
|---|---|
| INVESTIGAT | OR STATEMENT |
| I have read the Master Protocol, current sub-protocol, including all appendices, and I agree that is contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated. | |
| I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Vir Biotechnology, Inc. I will discuss this material with them to ensure they are fully informed about the drugs and the study. | |
| Principal Investigator Printed Name | Signature |
| | Date |

# PROTOCOL AMENDMENT 3 (26 JANUARY 2024) SUMMARY OF CHANGES TABLE

**Table 1:** Protocol Document History

| Document | Date |
|-------------------|-----------------|
| Amendment 3 | 26 January 2024 |
| Amendment 2 | 11 October 2022 |
| Amendment 1 | 16 May 2022 |
| Original Protocol | 01 April 2022 |

Summaries of changes for previous amendments are provided in Section 10.5.

**Table 2:** Protocol Amendment 3 Summary of Changes

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 1.1. Synopsis (Number of Participants), 4.1.1. Number of Participants, 9.2. Sample Size Determination, 9.5. Interim Analysis | Clarified that floater participants may be added at any time at Sponsor's discretion. As a result of this clarification, language in Section 9.5 (Interim Analysis) was updated for consistency | To clarify when floater participants can be added during the study |
| 2.3.1. Risk Assessment | Updated risk information for hypersensitivity reactions and immunogenicity for VIR-3434 | To provide updated risk assessment information for VIR-3434 per the most recent IB |
| 4.1.3. NRTI Treatment | Clarified that confirmatory test for HBV DNA > 20,000 IU/mL should occur no later than 7 calendar days after initial result is received. Also clarified that central laboratory testing is preferred, but local laboratory results will be accepted if it is not feasible to collect central laboratory results in time. | To ensure retesting is done promptly for safety management of participants who may be recommended to start NRTI therapy in follow-up period |
| 5.1. Inclusion Criteria | Clarified that participants must have HBV DNA $\leq 2,000 \text{ IU/mL}$ and $> LLOQ$ to be eligible | Participants must have quantifiable HBV DNA to be eligible |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 7.2. Discontinuation of Study Intervention(s) | Added the following additional treatment discontinuation criteria: | This change was made to include additional criteria for treatment discontinuation and |
| | Serum ALT or aspartate aminotransferase (AST) > 3 × ULN with: | clarification for when the Investigator may<br>stop study intervention. This change was |
| | serum albumin <3.0g/dL or | previously made in Addendum France-1 of VIR-SHB1-V202 (THRIVE) Amendment 2, |
| | ascites, hepatic encephalopathy, or liver-related<br>symptoms (eg, severe fatigue, nausea, vomiting, right<br>upper quadrant pain in the absence of an alternative<br>medical explanation) | Version 3.0 in response to a request made by ANSM of France and is being added to VIR-SHB1-V202 (THRIVE) Amendment 3 to harmonize into a single global protocol. |
| | Also added study intervention may be discontinued in the occurrence of a condition that in the opinion of the Investigator significantly jeopardizes the wellbeing and safety of the participant. Investigator must promptly inform the Sponsor Medical Monitor if any such condition arises. | |
| 8.8. Pharmacokinetic Assessments | Clarified that PK assessments are exploratory and may<br>or may not be analyzed, and specific assays used for<br>these assessments may be changed at the Sponsor's<br>discretion based on emerging data | To allow for appropriate analyses of exploratory PK assessments based on emerging data |
| 10.2. Appendix 2: Clinical<br>Laboratory Tests, 10.7. Appendix 7:<br>Additional Assessments in<br>Participants That Experience ALT<br>Elevation Meeting ECI Criteria | Added serum phosphate to the protocol-required safety laboratory tests | To align with renal monitoring guidance in the Viread® SmPC. This change was previously made in Addendum-1 and Addendum France-1 of VIR-SHB1-V202 (THRIVE) Amendment 2, Version 3.0 and is being added to VIR-SHB1-V202 (THRIVE) Amendment 3 to harmonize into a single global protocol. |

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 10.2. Appendix 2: Clinical<br>Laboratory Tests | Added footnote to clarify creatinine clearance calculation for study visits where weight is not measured (creatinine clearance will be calculated using the value measured from the most recent study visit) | To provide further guidance for creatinine clearance calculation. This clarification was described in Protocol Administrative Letter 1 for VIR-SHBV1-V202 (THRIVE) Amendment 2, Version 3.0 and is being added to VIR-SHB1-V203 (THRIVE) Amendment 3 to harmonize into a single global protocol. |
| Entire document | Other administrative, formatting, and other minor changes | These changes were made to clarify, ensure consistency, provide up-to-date information, or rectify typographical errors. |

# TABLE OF CONTENTS

| INVESTIC | GATOR SIGNATURE PAGE | 2 |
|---|---|---|
| 1. | PROTOCOL SUMMARY | 11 |
| 1.1. | Synopsis | 11 |
| 1.2. | Study Schema | 14 |
| 1.3. | Schedule of Activities | 14 |
| 2. | INTRODUCTION | 15 |
| 2.1. | Background | 15 |
| 2.2. | Study Rationale | 16 |
| 2.3. | Benefit/Risk Assessment | 17 |
| 2.3.1. | Risk Assessment | 17 |
| 2.3.2. | Benefit Assessment | 21 |
| 2.3.3. | Overall Benefit Risk Conclusion | 21 |
| 3. | OBJECTIVES AND ENDPOINTS | 22 |
| 4. | STUDY DESIGN | 24 |
| 4.1. | Overall Study Design | 24 |
| 4.1.1. | Number of Participants | 24 |
| 4.1.2. | Intervention Groups and Duration | 24 |
| 4.1.2.1. | Intervention Groups | 24 |
| 4.1.2.2. | Cohort Initiation | 25 |
| 4.1.2.3. | Duration | 25 |
| 4.1.3. | NRTI Treatment | 25 |
| 4.1.4. | Long-term and Follow-Up Care | 26 |
| 4.2. | Scientific Rationale for Study Design | 26 |
| 4.2.1. | Rationale for VIR-3434 for the Treatment of Chronic HBV Infection | 26 |
| 4.2.2. | Rationale for VIR-2218 for the Treatment of Chronic HBV Infection | 28 |
| 4.2.3. | Rationale for VIR-3434 + VIR-2218 + TDF for the Treatment of Chronic HBV Infection | 29 |
| 4.3. | Justification for Dose | 29 |
| 4.3.1. | VIR-3434 Dose Selection | 29 |
| 4.3.2. | VIR-2218 Dose Selection | 31 |
| 4.3.3. | TDF Dose Selection | 32 |
| 4.4. | End of Study Definition | 32 |

| 5. | STUDY POPULATION | 33 |
|---|---|---|
| 5.1. | Inclusion Criteria | 33 |
| 5.2. | Exclusion Criteria | 34 |
| 5.3. | Lifestyle Considerations | 36 |
| 5.3.1. | Meals and Dietary Restrictions | 36 |
| 5.3.2. | Caffeine, Alcohol, and Tobacco | 36 |
| 5.3.3. | Activity | 36 |
| 5.4. | Screen Failures | 36 |
| 6. | STUDY INTERVENTION(S) AND CONCOMITANT THERAPY | 37 |
| 6.1. | Study Intervention(s) Administered | 37 |
| 6.2. | Preparation, Handling, Storage, and Accountability | 38 |
| 6.3. | Randomization and Blinding | 38 |
| 6.4. | Study Intervention Compliance | 38 |
| 6.5. | Dose Modification | 38 |
| 6.5.1. | Dose Modifications for TDF | 38 |
| 6.6. | Concomitant Therapy | 38 |
| 6.6.1. | Concomitant Therapy Not Permitted During the Study | 38 |
| 7. | DISCONTINUATION OF STUDY, STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 40 |
| 7.1. | Study Stopping Rules | 40 |
| 7.2. | Discontinuation of Study Intervention(s) | 40 |
| 7.3. | Participant Discontinuation/Withdrawal from the Study | 41 |
| 7.4. | Replacement of Participants | 41 |
| 7.5. | Lost to Follow-up | 41 |
| 8. | STUDY ASSESSMENTS AND PROCEDURES | 41 |
| 8.1. | Screening Period | 41 |
| 8.2. | Efficacy Assessments | 41 |
| 8.3. | Safety Assessments | 41 |
| 8.3.1. | Physical Examinations | 41 |
| 8.3.2. | Vital Signs | 41 |
| 8.3.3. | Clinical Safety Laboratory Tests | 41 |
| 8.3.4. | Pregnancy Testing | 42 |
| 8.3.5. | Local Tolerability | 42 |

| 8.4. | Assessment of Viral Parameters, Antiviral Activity, and Resistance Surveillance | 42 |
|---|---|---|
| 8.5. | CCI | 42 |
| 8.6. | Exploratory Assessments | 42 |
| 8.6.1. | Exploratory Analysis Samples | 42 |
| 8.6.2. | CCI | 42 |
| 8.6.2.1. | CCI | 43 |
| 8.6.2.2. | CCI | 43 |
| 8.6.2.3. | CCI | 43 |
| 8.6.3. | CCI | 43 |
| 8.7. | Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Safety Reporting | 43 |
| 8.7.1. | Time Period and Frequency for Collecting AE and SAE Information | 43 |
| 8.7.2. | Follow-up of AEs and SAEs | 43 |
| 8.7.3. | Regulatory Reporting Requirements for SAEs. | 43 |
| 8.7.4. | Adverse Events of Interest | 43 |
| 8.7.5. | Clinical Laboratory Abnormalities and Other Abnormal Assessments as AEs or SAEs | 43 |
| 8.7.6. | Laboratory Events of Clinical Interest | 44 |
| 8.7.7. | Special Situation Reports | 44 |
| 8.7.7.1. | Pregnancy | 44 |
| 8.8. | Pharmacokinetic Assessments | 44 |
| 8.9. | Immunogenicity Assessments | 44 |
| 8.10. | Electrocardiogram | 44 |
| 8.11. | Liver Elastography (eg, FibroScan) | 44 |
| 9. | STATISTICAL CONSIDERATIONS | 45 |
| 9.1. | Statistical Hypotheses | 45 |
| 9.2. | Sample Size Determination | 45 |
| 9.3. | Analysis Sets | 46 |
| 9.4. | Statistical Analyses | 46 |
| 9.4.1. | General Considerations | 46 |
| 9.4.2. | Primary Endpoint(s) Analysis | 46 |
| 9.4.2.1. | Target Population. | 46 |

| 9.4.2.2. | Population Level Summary | 46 |
|---|---|---|
| 9.4.3. | Secondary Endpoint(s) Analysis | 47 |
| 9.4.4. | Exploratory Endpoint(s) Analysis | 47 |
| 9.4.5. | Missing Data | 47 |
| 9.4.6. | Other Safety Analyses | 47 |
| 9.5. | Interim Analysis | 47 |
| 9.6. | Pharmacokinetic Analyses | 48 |
| 9.7. | Immunogenicity Analyses | 48 |
| 10. | SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 49 |
| 10.1. | Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 49 |
| 10.1.1. | Regulatory and Ethical Considerations | 49 |
| 10.1.2. | Financial Disclosure | 49 |
| 10.1.3. | Informed Consent Process | 49 |
| 10.1.4. | Data Protection | 49 |
| 10.1.5. | Confidentiality | 49 |
| 10.1.6. | Committees Structure | 49 |
| 10.1.6.1. | Liver Flare Adjudication Committee (LFAC) | 49 |
| 10.1.7. | Dissemination of Clinical Study Data | 49 |
| 10.1.8. | Data Quality Assurance | 49 |
| 10.1.9. | Source Documents | 49 |
| 10.1.10. | Electronic Case Report Forms (eCRF) | 49 |
| 10.1.11. | Study and Site Start and Closure | 50 |
| 10.1.12. | Publication Policy | 50 |
| 10.2. | Appendix 2: Clinical Laboratory Tests | 51 |
| 10.3. | Appendix 3: AEs, SAEs, SSRs and AEIs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting | 53 |
| 10.4. | Appendix 4: List Abbreviations and Definitions of Terms | 54 |
| 10.5. | Appendix 5: Summaries of Changes for Previous Protocol Amendments | 56 |
| 10.6. | Appendix 6: Contraceptive and Barrier Guidance | 62 |
| 10.7. | Appendix 7: Additional Assessments in Participants That Experience ALT Elevation Meeting ECI Criteria | 64 |
| 10.8. | Appendix 8: Anaphylaxis, Cytokine Release Syndrome, And Immune<br>Complex Disease Supportive Measures | 66 |

| J | -, | |
|---|---|---|
| 10.9. | Appendix 9: Schedule of Activities | 68 |
| 11. | REFERENCES | 80 |
| | LIST OF TABLES | |
| Table 1: | Protocol Document History | 3 |
| Table 2: | Protocol Amendment 3 Summary of Changes | 3 |
| Table 3: | Intervention Groups | 24 |
| Table 4: | Study Intervention (s) Administered | 37 |
| Table 5: | Study Arm(s) | 37 |
| Table 6: | Protocol-Required Safety Laboratory Tests | 51 |
| Table 7: | Assessments in Participants That Experience ALT Elevation Meeting ECI Criteria | 64 |
| Table 8: | Schedule of Activities: Cohort 1b | 68 |
| Table 9: | Schedule of Activities: Cohort 2b | 72 |
| Table 10: | Schedule of Activities for Follow-Up Period for all Cohorts | 77 |
| | LIST OF FIGURES | |
| Figure 1: | Study Schema | 14 |
| Figure 2: | Dosing Scheme by Cohort | 14 |
| Figure 3: | Stages of Chronic HBV Infection | 15 |
| Figure 4: | VIR-3434 Observed and Projected Mean Concentration Profile in Healthy Volunteers in the Absence of HBsAg | 30 |

### 1. PROTOCOL SUMMARY

# 1.1. Synopsis

#### **Study Title**

A Phase 2 Study Evaluating the Efficacy and Safety of VIR-3434 and/or VIR-2218 containing regimens in HBeAg-negative Participants with Low Viral Burden of Chronic Hepatitis B Infection (THRIVE)

#### **Brief Title**

A Phase 2 Study to Evaluate VIR-3434 and/or VIR-2218 Containing Regimens for Treatment of Chronic Hepatitis B Infection

## **Background and Rationale**

Chronic HBV infection remains an important global public health problem with significant morbidity and mortality (Trepo 2014). Chronic HBV infection is a dynamic process characterized by the interplay of viral replication and the host immune response. Patients can be divided into different stages of the disease based on the levels of Hepatitis B e antigen (HBeAg), HBV DNA, alanine aminotransferase (ALT), and liver inflammation (EASL 2017; Sarin 2015; Terrault 2018).

Among the 300 million patients infected chronically with HBV, those who are HBeAg-negative represent the largest subgroup. These patients range from being inactive carriers to having chronic active hepatitis that can progress to serious liver complications including hepatocellular carcinoma (HCC). Inactive carriers are HBeAg-negative and anti-HBe-positive with persistently low levels of HBV DNA (≤ 2,000 IU/mL) and normal ALT maintained for at least 1 year. These patients have a good long-term prognosis with low rates of histological progression, low risk of cirrhosis or HCC, and high rates of long-term Hepatitis B surface antigen (HBsAg) clearance (EASL 2017; Invernizzi 2016; Terrault 2018; Yeo 2020). Inactive carriers lack indications for currently available treatments aimed at HBV DNA suppression, but they may be most likely to achieve functional cure, thereby becoming non-infectious with a lower risk of disease reactivation.

VIR-3434 is a monoclonal antibody targeting HBsAg with multiple potential mechanisms of action including strong neutralizing activity and enhanced immunologic activity due to Fc domain engineering. VIR-2218 is small interfering RNA (siRNA) that targets all HBV RNA transcripts and is associated with substantial reductions in HBsAg in patients with chronic HBV infection. VIR-3434 and TDF with or without VIR-2218 has the potential to achieve a functional cure of chronic HBV infection.

# **Primary and Secondary Objectives and Endpoints:**

The objectives and endpoints specific to this sub-protocol are listed in the table.

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of VIR-3434 and<br>tenofovir disoproxil fumarate (TDF) with or<br>without VIR-2218 | Proportion of participants achieving<br>suppression of HBV DNA (< LLOQ) with<br>HBsAg loss (< 0.05 IU/mL) at the end of<br>treatment <sup>a</sup> |
| Secondary | |
| <ul> <li>In addition to the Master Protocol,</li> <li>To assess the effect of VIR-3434 and TDF with or without VIR-2218 on HBV DNA</li> <li>To assess the effect of VIR-3434 and TDF with or without VIR-2218 on HBsAg</li> <li>To assess the immunogenicity of VIR-3434</li> </ul> | In addition to the Master Protocol secondary endpoints 1-8, 9. Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) after discontinuation of all treatment a. at 24 weeks b. at 48 weeks 10. Proportion of participants achieving HBsAg loss (< 0.05 IU/mL) a. at end of treatment b. at 24 weeks post-end of treatment 11. Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) after discontinuation of all treatment a. at 24 weeks b. at 48 weeks 12. Incidence and titers of anti-drug antibodies (ADA; if applicable) to VIR-3434 13. Mean change in serum HBsAg level from baseline across timepoints in the study 14. Proportion of participants achieving HBV DNA (< LLOQ) |

<sup>&</sup>lt;sup>a</sup> End of treatment as defined in SOA

#### **Overall Study Design**

This sub-protocol (THRIVE) should be read and conducted in conjunction with the PREVAIL Master Protocol. The Master Protocol provides a study framework: study outline, populations, common objectives and endpoints, common inclusion and exclusion criteria, statistical methodology, assessments and planned analyses for all sub-protocols. This sub-protocol is a Phase 2, multi-center, open-label study designed to evaluate the safety and efficacy of regimens containing VIR-3434 and NRTI with or without VIR-2218 in non-cirrhotic adult participants with low viral burden of chronic HBV infection.

### **Brief Summary**

This sub-protocol is intended to evaluate 24- to 48- week regimens of VIR-3434 and TDF with or without VIR-2218 in participants with chronic HBV infection. Study population IV as defined in the Master Protocol (and table below) as participants that are HBeAg negative with low HBV DNA ( $\leq 2,000 \text{ IU/mL}$ ) and ALT levels  $\leq$  ULN within the 1-year period prior to screening will be included in this sub-protocol.

| Master Protocol Population | HBeAg Status | HBV DNA Level | ALT Level |
|----------------------------|--------------|---------------|-----------|
| IV | Negative | ≤ 2,000 IU/mL | ≤ULN |

## **Number of Participants**

Up to 60 participants are planned to enroll in this sub-protocol. Cohorts 1b and 2b will each enroll approximately 15 participants initially. Additionally, up to 30 floater participants may be added to any of the cohorts in the sub-protocol at any time at Sponsor's discretion.

#### **Intervention Groups and Duration**

| Cohort | Study<br>Intervention | Dose | Route | Number of<br>Doses | Frequency of Dosing |
|---|---|---|---|---|---|
| 1b | VIR-3434 | 300 mg | SC | 12 | Every 4 weeks |
| | TDF | 300 mg <sup>a</sup> | Oral | 308 | Every day |
| 2b | VIR-3434 | 300 mg | SC | 12 | Every 4 weeks |
| | VIR-2218 | 200 mg | SC | 12 | Every 4 weeks |
| | TDF | 300 mg <sup>a</sup> | Oral | 308 | Every day |

<sup>&</sup>lt;sup>a</sup> Tenofovir disoproxil fumarate (TDF) dose will be 300 mg per label. Supply outside the United States may be tenofovir disoproxil (TD) 245 mg per label

The total duration in the study for all participants will be up to 100 weeks. This includes the Screening Period up to 56 days (8 weeks), the Treatment Period of 44 weeks, and a Follow-Up Period of 48 weeks.

# **Liver Flare Adjudication Committee (LFAC):**

The Liver Flare Adjudication Committee (LFAC) will provide hepatic safety oversight by performing periodic reviews of data pertaining to participants who meet certain prespecified criteria for ALT elevations (Section 8.7.6). The LFAC membership composition, laboratory criteria to trigger patient case evaluation by the LFAC, and data review requirements are described in detail in the LFAC Charter. (See Section 10.1.6.1)

# 1.2. Study Schema

Eligible participants will be enrolled via an interactive response technology (IRT) into 1 of the open cohorts. The overall study scheme is shown in Figure 1, and the dosing scheme for all cohorts are shown in Figure 2. The SOA for Cohorts 1b and 2b are provided in Table 8 and Table 9. Table 10 shows the SOA for the Follow-Up Period.

Figure 1: Study Schema



Figure 2: Dosing Scheme by Cohort



FU: Follow-Up; EOT: End of Treatment; Q4W: Every 4 weeks; TDF: Tenofovir disoproxil fumarate; HBsAg = Hepatitis B surface antigen; HBV DNA = Hepatitis B virus DNA; LLOQ = lower limit of quantitation See Section 4.1 for more details.

# 1.3. Schedule of Activities

Schedules of activities (SOA) are provided in Section 10.9.

## 2. INTRODUCTION

This sub-protocol should be read and conducted in conjunction with the PREVAIL Master Protocol (VIR-MHB1-V200).

# 2.1. Background

Chronic HBV infection remains an important global public health problem with significant morbidity and mortality (Trepo 2014). Chronic HBV infection is a dynamic process characterized by the interplay of viral replication and the host immune response. Patients can be divided into different stages of the disease based on the levels of Hepatitis B e antigen (HBeAg), Hepatitis B virus (HBV) DNA, ALT, and liver inflammation (EASL 2017; Sarin 2015; Terrault 2018).

Chronic HBV infection is a dynamic process and depends on the relationship between viral replication and host immune responses. Patients may oscillate between different phases of the disease, and serial monitoring of biomarkers such as HBV DNA, ALT, and HBV antigens helps determine the natural history of the disease. (Figure 3)

Figure 3: Stages of Chronic HBV Infection



Among the 300 million patients infected chronically with HBV, those who are HBeAg-negative represent the largest subgroup. These patients range from being immune inactive (also referred to as "inactive carriers" or "inactive hepatitis") to having chronic active hepatitis that can progress to serious liver complications including hepatocellular carcinoma (HCC). Inactive carriers are HBeAg-negative and anti-HBe-positive with persistently low levels of HBV DNA (< 2,000 IU/mL) and normal ALT maintained for at least 1 year. These patients have a good long-term prognosis with low rates of histological progression, low risk of cirrhosis or HCC, and high rates of long-term HBsAg clearance (EASL 2017; Invernizzi 2016; Terrault 2018; Yeo 2020). Inactive carriers lack indications for currently available treatments aimed at HBV DNA suppression, but they may be most likely to achieve functional cure, thereby becoming non-infectious with a lower risk of disease reactivation.

# 2.2. Study Rationale

VIR-3434 is a monoclonal antibody (mAb) targeting Hepatitis B surface antigen (HBsAg) with multiple potential mechanisms of action, including strong neutralizing activity and enhanced immunologic activity due to Fc domain engineering. In patients with chronic HBV infection, prior studies have shown that restoration of HBV-specific CD8+ T cell function by PD-1 blockade in immune inactive patients is linked to T cell differentiation (Bengsch 2014). Reports from this study suggest that the potential to revive HBV-specific T cells in an immune inactive population may be feasible with VIR-3434's proposed mechanism as a vaccinal mAb with T cell engagement activity. VIR-2218 is a siRNA that is associated with substantial reductions in HBsAg in patients with chronic HBV infection. VIR-3434 and an NRTI, with or without VIR-2218, have the potential to achieve a functional cure of chronic HBV infection.

See Section 4.2 for additional scientific rationale for the different investigational regimens in this sub-protocol.

# 2.3. Benefit/Risk Assessment

Detailed information about the known and potential benefits and risks of VIR-2218 and VIR-3434 may be found in the respective Investigator's Brochures (IBs).

# 2.3.1. Risk Assessment

| Potential Risk of Clinical Summary of Data/Rationale for Risk Significance | | Mitigation Strategy |
|---|---|---|
| | Study Intervention: VIR-2218 | |
| Injection site reactions (ISRs) | Based on available preliminary clinical data from studies VIR-2218-1001 and VIR-2218-1006, ISRs are a recognized risk of subcutaneous (SC) administered siRNA therapies and are typically transient. | Participants are monitored for local tolerability after injection and all AEs will be collected to reflect any ISRs that may be reported. Routine safety monitoring and reporting procedures are in place to provide safety overview. |
| Immunogenicity: Immunogenicity is a potential risk associated with siRNA molecules. In general, the development of anti-drug antibodies (ADA) may impact safety, efficacy, or both. | Immunogenicity data from Parts B/C of the VIR-2218-1001 study indicated a low immunogenicity risk based on all confirmed participants yielding negative titers. | While there were no apparent clinical consequences related to the presence of VIR-2218 ADA, immunogenicity will continue to be assessed in Parts D/F of study VIR-2218-1001. |
| Liver function test abnormalities: VIR-2218 is targeted for delivery to the liver, and transient transaminase elevations have been observed with SC administration with other GalNAc-conjugated siRNA therapeutics. | Based on available preliminary clinical data from studies VIR-2218-1001 and VIR-2218-1006, minor ALT elevations (Grade 1 or Grade 2) have been observed in participants receiving VIR-2218 monotherapy. However, none of the participants met Hy's law and the majority resolved the ALT elevations by the end of treatment. | Monitoring of liver function is recommended. In addition, ALT flares in chronic HBV patients may be a sign of restoration of HBV-targeted immunity, therefore close monitoring of liver function and HBV-viral parameters may be warranted. Low probability: Events of Clinical Interest (ECI) defined as ALT elevations >3x ULN, must be reported within 5 business days of Investigator notification. The Sponsor will monitor ECI and an independent Liver Flare Adjudication Committee (LFAC) reviews the liver safety and assesses etiology to recommend changes in study conduct. |

| Potential Risk of Clinical Summary of Data/Rationale for Risk Significance | | Mitigation Strategy |
|---|---|---|
| Probability of significant non-target mediated toxicity: Hypersensitivity reactions (including injection site reactions [ISRs] and anaphylaxis): Hypersensitivity reactions (including ISRs and anaphylaxis), which may be severe or life-threatening, are a potential risk associated with the mAb class. The distinct risk of developing such conditions after dosing with VIR-3434 is unknown. | Based on data from completed study VIR-3434-1002 and available preliminary data from ongoing study VIR-2218-1006, VIR-3434 has been generally well tolerated in healthy participants and in participants with chronic HBV infection. ISRs that are Grade 1 or 2 in severity and transient have been observed with SC administration of VIR-3434. Most ISRs were considered unrelated to VIR-3434. | Low probability: participants will be closely monitored to evaluate any patterns of non-target mediated toxicity. Participants are monitored for local tolerability after injection and all AEs will be collected to reflect any hypersensitivity reactions that may be reported. Routine safety monitoring and reporting procedures are in place to provide safety overview. |
| Immunogenicity: Immunogenicity is a potential risk associated with the mAb class. VIR-3434 is a human immunoglobulin G (IgG) mAb; therefore, the development of ADA may impact its safety, efficacy, or both. | In completed study VIR-3434-1002, there was no observable effect of ADA on PK, safety, and efficacy in the participants with treatment-emergent ADA. | Immunogenicity data will continue to be monitored and assessed in relation to associated VIR-3434 PK and clinical safety measures. |
| Potential target-mediated risks: immune complex disease and hepatotoxicity due to the elimination of infected hepatocytes via cytotoxic T-cells induced via a vaccinal effect. As no or only low levels of HBsAg is detected on the surface of infected hepatocytes, antibody-dependent cellular cytotoxicity (ADCC)/antibody-dependent cellular phagocytosis (ADCP)-mediated elimination of hepatocytes is possible but unlikely to occur. | In study VIR-3434-1002, single doses up to 300 mg were well tolerated. No clinically significant changes in laboratory parameters were observed, and no participant developed clinical or laboratory evidence of immune complex disease. These preliminary results are consistent with prior clinical experience supporting the safety of anti-HBsAg mAb. HBV-AB <sup>XTL</sup> , a mixture of two anti-HBsAg monoclonal antibodies, was evaluated at doses up to 80 mg administered weekly for 4 doses in patients with baseline HBsAg ranging from approximately 20 to | Low probability: participants will be closely monitored to evaluate any patterns of non-target mediated toxicity. |

| Potential Risk of Clinical<br>Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | 80,000 IU/mL, and no signs of immune complex disease or hepatotoxicity were observed (Galun 2002). Additionally, several studies have evaluated the use of hepatitis B immune globulin (HBIG) in patients with chronic HBV infection and reported favorable safety and tolerability (Perrillo 2013, Reed 1973, Tsuge 2016). In the largest study, 64 patients with baseline HBsAg ranging from 0.09 to 11,214 IU/mL (mean 1,965 IU/mL) received HBIG therapy for multiple weeks, and no clinical manifestations of immune complex disease or other safety concerns were observed (Perrillo 2013). | |
| | Study Intervention: VIR-3434 + VIR-2218 | 3 + TDF |
| Hepatotoxicity | The combination of these study interventions may result in hepatotoxicity (eg, elevated ALT). Based on available preliminary clinical data from ongoing studies VIR-2218-1001 and VIR-2218-1006 and completed study VIR-3434-1002: VIR-2218 or VIR-3434 monotherapy in virally suppressed participants have resulted in minor ALT elevations (Grade 1 or Grade 2). However, none of the participants met Hy's law, and the majority of ALT elevations resolved after the end of treatment. | Addition of NRTI (TDF [tenofovir disoproxil fumarate]) to the treatment regimen to suppress viral replication Excluding patients with significant fibrosis or cirrhosis, significant chronic liver disease (except HBV infection), history of hepatic decompensation. Routine safety monitoring and reporting procedures ECI; defined as ALT elevations >3x ULN must be reported within 5 business days of Investigator notification. Sponsor monitors ECI and an independent Liver Flare Adjudication Committee (LFAC) reviews the liver safety and assesses etiology to recommend changes in study conduct Stopping criteria for study interventions have been provided in Section 7.1. |

| Potential Risk of Clinical<br>Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Injection site reactions | Combination of VIR-3434 +/- VIR-2218 may result in ISRs such as injection site pain, bruising, itching, rash. In the completed VIR-3434-1002 study and ongoing VIR-2218-1001 and VIR-2218-1006 studies, these interventions alone on or in combination have resulted in ISRs Grade 1 or 2 in severity that usually resolve within a few days to weeks. There is no potential cumulative risk for the combination intervention of VIR-3434 + VIR-2218. | Participants are monitored for local tolerability after injection and all AEs will be collected to reflect any ISRs that may be reported. Routine safety monitoring and reporting procedures are in place to provide safety overview. |

#### 2.3.2. Benefit Assessment

Single doses of VIR-2218 up to 900 mg in healthy volunteers and up to 6 doses of up to 200 mg administered every 4 weeks (ie, the highest dose tested) in participants with chronic HBV infection were well tolerated and exhibited safety profiles supportive of continued clinical development (VIR-2218 Investigator's Brochure). Regardless of hepatitis B e antigen (HBeAg) status, VIR-2218 was associated with a -1.96 log10 IU/mL mean decrease in HBsAg after 6 every 4-week (Q4W) doses (Lim 2022).

VIR-3434 has the potential to further reduce HBsAg, inhibit the intrahepatic spread of HBV via entry inhibition, eliminate infected hepatocytes, and stimulate an adaptive immune response against HBV. Lower HBsAg levels that may be achieved by lead-in or concomitant administration of VIR-2218 have the potential to augment the effects of VIR-3434 and achieve a functional cure of chronic HBV infection. Additionally, multiple-dose regimens of VIR-3434 may produce rapid and sustained reductions of HBsAg in the absence of VIR-2218 and potentially achieve functional cure of chronic HBV infection as monotherapy.

In the ongoing VIR-2218-1001 study, monotherapy with 6 doses of VIR-2218 is being evaluated in virally suppressed (on NRTI) participants with chronic HBV infection. Preliminary safety and tolerability data suggest VIR-2218 monotherapy was generally well-tolerated (Yuen 2021). Additionally, substantial sustained reductions in HBsAg were observed, compared to 2 doses of VIR-2218 in Parts B-C (Lim 2022). In this sub-protocol, it is hypothesized that the addition of VIR-3434 to VIR-2218 will lead to higher rates of HBsAg loss and functional cure.

#### 2.3.3. Overall Benefit Risk Conclusion

The patient population in this study will have low level viremia and liver inflammation. This study will provide information on the safety, tolerability, and efficacy of VIR-3434 and NRTI (TDF) in combination with VIR-2218. The study is designed to test the hypothesis that regimens containing VIR-3434 and TDF with or without VIR-2218 may lead to a functional cure of chronic HBV infection by reducing HBsAg and stimulating a host immune response. Compared to the current standard of care, the regimens in this study offer the potential benefits of finite duration, pangenotypic activity, and the potential to achieve functional cure, which may be associated with a reduction in serious HBV-associated sequelae such as cirrhosis, liver failure, HCC, or death.

The mechanistic rationale, together with available clinical data, supports a favorable risk-benefit profile for evaluation of regimens containing VIR-3434, TDF, and/or VIR-2218 in patients with chronic HBV infection.

# 3. OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of VIR-3434 and TDF with or without VIR-2218 | Proportion of participants achieving<br>suppression of HBV DNA (< LLOQ) with<br>HBsAg loss (< 0.05 IU/mL) at the end of<br>treatment <sup>a</sup> |
| Secondary | |
| <ul> <li>In addition to the Master Protocol objectives,</li> <li>To assess the effect of VIR-3434 and TDF with or without VIR-2218 on HBV DNA</li> <li>To assess the effect of VIR-3434 and TDF with or without VIR-2218 on HBsAg</li> <li>To assess the immunogenicity of VIR-3434</li> </ul> | In addition to the Master Protocol secondary endpoints 1-8, 9. Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) after discontinuation of all treatment a. at 24 weeks b. at 48 weeks 10. Proportion of participants achieving HBsAg loss (< 0.05 IU/mL) a. at end of treatment b. at 24 weeks post-end of treatment <sup>a</sup> 11. Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) after discontinuation of all treatment a. at 24 weeks b. at 48 weeks 12. Incidence and titers of ADA (if applicable) to VIR-3434 13. Mean change in serum HBsAg level from baseline across timepoints in the study 14. Proportion of participants achieving HBV DNA (< LLOQ) |

| Objectives | | Endpoints |
|---|---|---|
| Ex | Exploratory | |
| | addition to the Master Protocol objectives. To evaluate proportion of participants meeting criteria for nucleos(t)ide reverse transcriptase inhibitor (NRTI) treatment after discontinuation of all treatments To assess the effect of the VIR-3434 and TDF with or without VIR-2218 on HBV DNA To characterize the pharmacokinetics (PK) of VIR-3434 To characterize the PK of VIR-2218 (for cohorts with VIR-2218) To assess the immunogenicity of VIR-2218 (for cohorts with VIR-2218) | <ul> <li>In addition to the Master Protocol exploratory endpoints 1-6.</li> <li>7. Proportion of participants meeting criteria for NRTI treatment in Follow-Up Period</li> <li>8. HBV DNA levels and change from baseline across timepoints in the study</li> <li>9. Nadir and maximum change of HBV DNA levels from baseline in the study</li> <li>10. VIR-3434 PK parameters</li> <li>11. VIR-2218 PK parameters (for cohorts with VIR-2218)</li> <li>12. Incidence and titers of ADA (if applicable) to VIR-2218 (for cohorts with VIR-2218)</li> <li>13. Proportion of participants with virological</li> </ul> |
| • | To assess the effect of duration of treatment of VIR-3434 and TDF with or without VIR-2218 | 13. Proportion of participants with virological relapse (defined as either (1) an increase of |
| • | To assess potential virological relapse | ≥ 1 log <sub>10</sub> HBV DNA IU/mL above nadir for at least 2 consecutive visits OR (2) quantifiable HBV DNA of ≥ 1 log <sub>10</sub> IU/mL above LLOQ for at least 2 consecutive visits after being < LLOQ) |

<sup>&</sup>lt;sup>a</sup> End of treatment as defined in SOA

### 4. STUDY DESIGN

# 4.1. Overall Study Design

The THRIVE sub-protocol should be read and conducted in conjunction with the PREVAIL Master Protocol. The Master Protocol provides a study framework: study outline, populations, common objectives and endpoints, common inclusion and exclusion criteria, statistical methodology, assessments and planned analyses for all sub-protocols. THRIVE is a Phase 2, multi-center, open-label study designed to evaluate the safety and efficacy of regimens containing VIR-3434 and NRTI with or without VIR-2218 in non-cirrhotic adult participants with low viremic burden of chronic HBV infection currently not on treatment. The study is planned to be conducted at multiple clinical investigative sites globally.

The THRIVE sub-protocol is intended to evaluate up to 48-week regimens of VIR-3434 in combination with tenofovir disoproxil fumarate (TDF) with or without VIR-2218 in participants with chronic HBV infection. Study population IV as defined in the Master Protocol (and table) that are HBeAg negative with low HBV DNA ( $\leq 2,000 \text{ IU/mL}$ ) and ALT levels  $\leq$  ULN within the 1-year period prior to screening will be included in this sub-protocol.

| Master Protocol Population | HBeAg Status | HBV DNA Level | ALT Level |
|----------------------------|--------------|---------------|-----------|
| IV | Negative | ≤ 2,000 IU/mL | ≤ULN |

# 4.1.1. Number of Participants

Up to 60 participants are planned to enroll in this sub-protocol. Cohorts 1b and 2b will each enroll approximately 15 participants initially. An additional 30 participants may be added to any of the cohorts in this sub-protocol at any time at Sponsor's discretion.

# 4.1.2. Intervention Groups and Duration

#### 4.1.2.1. Intervention Groups

There are 2 cohorts planned in this sub-protocol (Table 3).

**Table 3:** Intervention Groups

| Cohort | Study intervention | Dose | Route | Number of<br>Doses | Frequency of Dosing |
|---|---|---|---|---|---|
| 11. | VIR-3434 | 300 mg | SC | 12 | Every 4 weeks |
| 1b | TDF | 300 mg <sup>a</sup> | Oral | 308 | Every day |
| | VIR-3434 | 300 mg | SC | 12 | Every 4 weeks |
| 2b | VIR-2218 | 200 mg | SC | 12 | Every 4 weeks |
| | TDF | 300 mg <sup>a</sup> | Oral | 308 | Every day |

<sup>&</sup>lt;sup>a</sup> Tenofovir disoproxil fumarate (TDF) dose will be 300 mg per label. Supply outside the United States may be Tenofovir disoproxil (TD) and the corresponding dose will be 245 mg per label.

#### 4.1.2.2. Cohort Initiation

Cohorts in this study may be enrolled in parallel. Cohorts may be opened, closed, or discontinued at the Sponsor's discretion.

#### **4.1.2.3. Duration**

The total duration for participants in Cohorts 1b and 2b will be up to 100 weeks inclusive of the Screening Period, Treatment Period, and Follow-Up Period.

## 4.1.2.3.1. Screening Period

The Screening Period for all participants will be up to 56 days (8 weeks).

#### 4.1.2.3.2. Treatment Period

The Treatment Period will be 44 weeks for Cohorts 1b and 2b.

## 4.1.2.3.3. Follow-Up Period

Once participants complete the Treatment Period per their respective cohort, they will enter the Follow-Up Period. The maximum duration of the Follow-Up Period is 48 weeks after the last dose of the study intervention(s).

#### 4.1.3. NRTI Treatment

It is recommended that commercial NRTI therapy be reinitiated in participants at any time during the Follow-Up Period if they meet any of the following criteria:

- HBV DNA increase  $\geq 2 \log_{10} IU/mL$  within a 2-week period
- HBV DNA > 100,000 IU/mL at any Follow-Up Period visit (regardless of other biochemical parameters or ALT values)
- Confirmed increase of HBV DNA > 20,000 IU/mL (ie, at 2 consecutive collections, regardless of other biochemical parameters or ALT values)
  - Note: The repeat HBV DNA test should be performed as soon as possible and no later than 7 calendar days after the initial result is received. Central laboratory testing is preferred, but local laboratory results will be accepted if it is not feasible to collect central laboratory results in time.

- HBV DNA > 2,000 IU/mL concurrent with any of the following criteria at the same visit:
  - Confirmed total bilirubin > 2x ULN and ALT > ULN
  - Any sign of hepatic decompensation (including, but not limited to, confirmed increase in prothrombin time [PT] ≥ 2 or international normalized ratio [INR] ≥ 0.5 from baseline, jaundice, ascites, encephalopathy, etc)
  - ALT > 10x ULN
  - ALT > 2x ULN persisting for  $\ge 12$  consecutive weeks
  - ALT > 5x ULN persisting for  $\ge 4$  consecutive weeks
- Confirmed HBeAg seroreversion (ie, HBeAg positive after being HBeAg negative)
- Any other clinically significant event(s) warranting initiation of NRTI therapy in the opinion of the investigator after discussion with Sponsor

Participants who start NRTI therapy in the Follow-Up period should continue to be followed per the SOA for the Follow-Up Period (Table 10) through the Week 48 visit. Participants with HBV DNA increase  $\geq 2 \log_{10} IU/mL$  within a 2-week period should:

- return to the site for an unscheduled visit to measure HBV DNA levels and liver function tests as soon as possible after the investigator becoming aware of the HBV DNA increase
- continue returning weekly until HBV DNA levels stabilize (do not increase ≥ 1 log<sub>10</sub> IU/mL over 4-week period or start decreasing for at least 2 consecutive visits) after which they should continue per the SOA for the Follow-Up Period

If any unscheduled visits needed as outlined above coincide with an existing visit per the Follow-Up Period SOA then the Follow-Up visit assessments should be conducted.

#### 4.1.4. Long-term and Follow-Up Care

Once a participant has completed the study, long-term care should be determined by the Investigator or primary treating physician based on local clinical guidelines.

# 4.2. Scientific Rationale for Study Design

### 4.2.1. Rationale for VIR-3434 for the Treatment of Chronic HBV Infection

VIR-3434 offers a novel strategy for the treatment of chronic HBV infection by neutralizing HBV viral and subviral particles through the targeting of HBsAg and inhibition of viral entry into hepatocytes. Additionally, the Fc region of VIR-3434 is engineered to increase binding affinity to the neonatal Fc receptor (FcRn) and promote the Fc-gamma receptor (Fc $\gamma$ R) binding profile towards the activating receptors. These modifications may prolong serum half-life, increase potency, and induce a "vaccinal" effect (the induction of antigen-specific T cell responses).

The normal serum half-life of IgG is approximately 21 days and regulated by a balance of FcRn-mediated endocytosis and recycling versus endosomal degradation. To produce a product with sustained activity against HBV, the well characterized LS modification (M428L and N434S) (Gaudinski 2018; Ko 2014; Zalevski 2010) was included in the Fc region of VIR-3434. The LS modification increases IgG1 binding to FcRn only at the acidic pH of the endosomal compartment thereby increasing IgG recycling back into circulation. Monoclonal antibodies containing the LS mutation have previously been studied in humans (Gaudinski 2018). For example, VRC01LS, a mAb against the CD4 binding site of the HIV-1 glycoprotein, was deemed safe and well tolerated at doses of 5 to 40 mg/kg IV and 5 mg/kg SC in healthy volunteers. No anti-drug antibodies (ADAs) were detected out to 48 weeks. VIR-3434 is similarly anticipated to have an extended half-life in humans, resulting in a prolonged duration of exposure. *In vitro* data for VIR-3434 suggests that the LS mutation is not anticipated to interfere with the additional Fc modifications described below.

The Fc region of VIR-3434 was also engineered to include a modification which modulates binding to human FcγRs by enhancing binding to the activating receptors FcγRIIa and FcγRIIIa, while diminishing binding to the inhibitory receptor FcγRIIb. This Fc modification is designed to enhance ADCP of HBsAg and HBV virions and antigen presentation and, as a result, promote the induction of T cell responses ("vaccinal effect"). The impact of similar modifications on mAb efficacy have been studied in a FcγR-humanized lymphoma mouse model. In this model, anti-CD20 antibodies promoted direct killing of tumor cells via engagement of FcγRIIIa on macrophages and monocytes. In addition, anti-CD20-immune complexes induced CD8+ T cell responses via FcγRIIa-dependent presentation of tumor antigens by dendritic cells. Overall, Fc-engineering of anti-CD20 antibodies to increase FcγRIIa and FcγRIIIa binding (GASDALIE mutation) had superior therapeutic activity (DiLillo 2015). Parallel reduction of binding to the inhibitory FcγRIIb has the potential to further augment this vaccinal effect (DiLillo 2015).

Available data regarding the use of HBsAg-directed antibodies in the treatment of patients with chronic HBV infection suggest that these molecules have the potential to reduce HBsAg levels while maintaining an acceptable safety and tolerability profile. GC1102, a fully human anti-HBsAg mAb in development for chronic HBV infection and prevention of recurrent HBV following liver transplantation, effectively lowered HBsAg by 2-3 log<sub>10</sub> IU/mL and was well tolerated in a Phase 1 study in patients with chronic HBV infection, with no evidence of serious sequelae such as immune complex disease (Lee 2018). HBV-AB<sup>XTL</sup> (HepeX-B), a mixture of two human anti-HBsAg mAbs, was administered to 27 patients with levels of HBsAg ranging from approximately 20 to 85,000 IU/mL. HBV-AB<sup>XTL</sup> was found to have a favorable safety and tolerability profile at doses up to 80 mg administered weekly for 4 doses, and no signs of immune complex disease or hepatotoxicity were reported (Galun 2002). Similarly, no adverse events were reported in two studies of chronic HBV patients receiving high doses of hepatitis B immune globulin (HBIG) to prevent re-infection following liver transplantation (Reed 1973; Tsuge 2016).

Clinical data from the oncology setting suggests that Fc engineering designed to enhance ADCC/ADCP, and antigen presentation may improve efficacy without compromising safety or tolerability (Im 2018). Margetuximab is a modified version of trastuzumab that has been approved by FDA for the treatment of HER2-positive carcinomas. Margetuximab contains modifications designed to enhance ADCC/ADCP and antigen presentation. Margetuximab was well tolerated in a first-in-human (FIH) Phase 1 study in patients with HER-2 positive carcinomas. Common toxicities were primarily ≤ Grade 2, including no evidence of cardiotoxicity (Bang 2017), which has been observed with the non-Fc modified parent mAb, trastuzumab, in late-stage clinical trials (Ponde 2016; Riccio 2016).

Taken together, these data suggest that mAbs that are Fc engineered to prolong serum half-life and optimize immune effector cell activity have the potential to improve the efficacy of therapeutic mAbs without compromising safety. VIR-3434 is predicted to decrease serum HBsAg, inhibit intrahepatic viral spread, eliminate infected hepatocytes, and stimulate HBV-specific immune responses. Therefore, VIR-3434 has the potential to achieve a functional cure of chronic HBV infection, with or without other agents such as VIR-2218 and an NRTI (TDF).

VIR-3434 has been evaluated in VIR-3434-1002 and is being evaluated in VIR-2218-1006 in participants with chronic HBV infection. Cohort 1b will assess the contribution of VIR-3434 to combination therapies and its potential to achieve functional cure in the absence of any other investigational agents. To assess participant responses and a potential vaccinal effect from VIR-3434, peripheral blood mononuclear cells (PBMCs) will be collected to perform evaluation of host cellular immune responses (eg, T cells) against HBV antigens.

#### 4.2.2. Rationale for VIR-2218 for the Treatment of Chronic HBV Infection

The use of siRNA offers a novel strategy for the treatment of chronic HBV infection. siRNAs are 19-21 base-pair RNA duplexes that exploit the endogenous RNA-interference pathway to enable sequence-specific RNA cleavage and degradation. One siRNA can have multiple antiviral effects, including degradation of the pgRNA, thus inhibiting viral replication, and degradation of all viral messenger RNA (mRNA) transcripts, thereby preventing expression of viral proteins. This may result in the return of a functional immune response directed against HBV, either alone or in combination with other therapies.

By contrast, NRTIs act at a distinct part of the viral life cycle and have a different mechanism of action than VIR-2218. NRTIs inhibit the HBV polymerase, blocking the reverse transcription of the viral pgRNA to viral DNA and preventing the production of infectious virions. NRTIs, however, do not directly impact the production of viral proteins such as HBsAg.

VIR-2218 is a GalNAc conjugated siRNA that targets all HBV viral RNA and thereby inhibiting production and secretion of virions and subviral particles. In the ongoing VIR-2218-1001 and VIR-2218-1006 studies, VIR-2218 alone and in combination with other agents (PEG-IFN or VIR-3434) has been shown to induce significant reductions in HBsAg levels in participants with chronic HBV infection.

Reduction of HBsAg-containing noninfectious subviral particles by VIR-2218 is considered an important differentiator from currently available treatments.

# 4.2.3. Rationale for VIR-3434 + VIR-2218 + TDF for the Treatment of Chronic HBV Infection

Emerging clinical data suggests that a combination of multiple therapeutic modalities may be necessary to achieve functional cure in the majority of chronic HBV patients (Revill 2019; Zoulim 2015). The excessive secretion of non-virion incorporated HBsAg in chronic HBV infection is thought to contribute to T and B cell dysfunction and to impair the host's ability to clear or control the virus (Bertoletti 2016; Burton 2018; Maini 2016). Therefore, development of functional cure is likely to require a reduction or elimination of HBsAg in conjunction with the induction of host immunity against the infection.

When administered individually, VIR-2218 and VIR-3434 are associated with substantial reductions in HBsAg in patients with chronic HBV infection (Gane 2021; Yuen 2021). The combination of VIR-2218 and VIR-3434 is thus anticipated to result in deep, sustained reductions in HBsAg. This is supported by AAV-HBV mouse model of chronic HBV infection, in which combination treatment with VIR-2218 and VIR-3434 was associated with marked reductions in HBsAg. Additionally, lower HBsAg levels achieved by prior or concomitant treatment with VIR-2218 may augment the effect of VIR-3434.

Reduction in HBsAg may also augment the potential immunologic effects of VIR-3434. The Fc modifications of VIR-3434 are designed to enhance ADCP of HBsAg and HBV virions and antigen presentation and, as a result, promote the induction of T cell responses. Given the putative impact of HBsAg on immune function, these potential effects of VIR-3434 may be enhanced in the setting of lower HBsAg, which can be achieved with lead-in and/or concurrent treatment with VIR-2218. Longer durations of VIR-3434 dosing may also enhance these effects.

The participant population included in this sub-protocol have a low viral burden and normal ALT, and are not indicated for treatment with NRTI. However, NRTIs such as TDF help reduce viral replication and thereby reduce the HBV DNA levels. Therefore, they are included as part of all regimens in this sub-protocol in addition to VIR-3434 to allow these participants with low HBV DNA levels to achieve HBV DNA < LLOQ along with VIR-3434 which has potential immune-modulatory effects to ultimately achieve sustained suppression of HBV DNA with or without HBsAg loss.

#### 4.3. Justification for Dose

#### 4.3.1. VIR-3434 Dose Selection

Available PK, safety, and antiviral activity from the VIR-3434-1002 and VIR-2218-1006 studies were considered for selection of the VIR-3434 dosing regimens.



VIR-3434 has a half-life ( $t_{1/2}$ ) of approximately 25 days, with measurable concentrations up to 24 weeks after a single SC dose of 90-900 mg in healthy volunteers (Gupta 2021). Dose-proportional increases in  $C_{max}$  and  $AUC_{inf}$  were observed across the SC dose range evaluated. A similar  $t_{1/2}$  was observed following a single IV injection of 3,000 mg. Nonparametric superposition was employed to predict the concentration time profile and PK exposures following 13 SC doses of VIR-3434 300 mg administered every 4 weeks. As seen in Figure 4, the projected  $C_{max}$  of 50  $\mu$ g/mL for this regimen would not exceed the observed  $C_{max}$  of a single 3,000 mg IV dose of 1,076  $\mu$ g/mL. Similarly, the projected AUC<sub>inf</sub> associated with this regimen (5,148 day\* $\mu$ g/mL) does not exceed the observed mean AUC<sub>inf</sub> of the 3,000 mg IV dose (11,842 day\* $\mu$ g/mL). Additionally, due to target-mediated drug disposition, the PK exposure in healthy volunteers is anticipated to be an overestimate compared to participants with chronic HBV infection, as VIR-3434 is expected to be eliminated more rapidly in the presence of HBsAg.

Figure 4: VIR-3434 Observed and Projected Mean Concentration Profile in Healthy Volunteers in the Absence of HBsAg



Mean concentration of VIR-3434 observed over time in healthy volunteers in VIR-3434-1002 administered single dose of VIR-3434 either 300 mg SC (green solid line) or 3000 mg IV (red solid line). The projected mean concentration profile of VIR-3434 following 13 doses of 300 mg SC administered every 4 weeks in the absence of HBsAg and assuming a 25-day half-life is depicted in blue.

Data from VIR-3434-1002 demonstrated that single doses of up to 300 mg VIR-3434 were generally well tolerated with no safety concerns in participants with chronic HBV infection. The majority of AEs were Grade 1 or 2. There were no study discontinuations due to AEs. In the ongoing VIR-2218-1006 study, combination regimens of VIR-3434 are being evaluated in participants with chronic HBV infection who are on NRTIs. No significant safety concerns have been identified to date for VIR-3434 up to 12 doses of up to 75 mg administered weekly. The cumulative exposure following 13 SC doses of VIR-3434 every 4 weeks at 300 mg is not anticipated to exceed the maximum exposure associated with a single dose of 3,000 mg administered IV in healthy volunteers.

Based on antiviral data in study VIR-3434-1002, VIR-3434 is associated with HBsAg reductions > 1 log<sub>10</sub> IU/mL in the majority of study participants following a single SC dose of 6 to 300 mg in a dose dependent manner (Agarwal 2021; Agarwal 2022). The 300 mg dose level was associated with the largest and most durable HBsAg reductions, with mean reductions from baseline of >2 log<sub>10</sub> at Week 4 and > 1.5 log<sub>10</sub> at Week 8. Repeat administration of VIR-3434 may enhance the reduction of HBsAg, increase the likelihood of eliciting the potential immunomodulatory effects of its Fc domain modifications, and prolong the duration of viral entry inhibition.

In summary, the observed PK, HBsAg kinetics and absence of safety signals in the ongoing single dose and multiple dose studies, along with the potential for multiple doses of VIR-3434 to further lower HBsAg, support the dose level, frequency, and duration of VIR-3434 regimens selected for this sub-protocol.

#### 4.3.2. VIR-2218 Dose Selection

Available safety, tolerability, antiviral activity, and pharmacokinetic data from Parts A-F of study VIR-2218-1001 were considered when selecting dose regimens for VIR-2218.

In Part A of the VIR-2218-1001 study, a single SC dose of VIR-2218 was administered to healthy volunteers over the dose range of 50 to 900 mg. In Parts B and C of the study, 2 doses of VIR-2218 given 4 weeks apart, ranging from 20 to 200 mg were administered to participants with chronic HBV infection. In healthy volunteers, VIR-2218 was absorbed after SC injection with a median  $T_{max}$  of 4-7 hours and was not measurable in plasma beyond 48 hours for any participant (Gupta 2021). Available PK data from HBV participants were similar to healthy adults. No accumulation of VIR-2218 in plasma was evident following a second dose of VIR-2218 administered 4 weeks apart in participants with chronic HBV infection.

In Cohort 2b of this study, VIR-2218 will be administered as a SC injection of 200 mg every 4 weeks for 12 doses. The duration of VIR-2218 treatment in each cohort was selected to ensure suppression of HBsAg by VIR-2218 for the entire duration of concomitant treatment with VIR-3434. Regimens containing varying durations up to 12 doses of 200 mg VIR-2218 administered every 4 weeks will be evaluated to assess the impact of more sustained HBsAg suppression on the outcome of functional cure.

The VIR-2218 dose level of 200 mg was selected based on results from Parts B and C of the VIR-2218-1001 study. In participants with chronic HBV infection, a regimen of 2 doses of VIR-2218 administered 4 weeks apart was associated with dose-dependent reductions in HBsAg across a dose range of 20-200 mg (Gane 2021; Lim 2022). The largest reductions in HBsAg were observed in the 200 mg cohort.

The VIR-2218 regimens selected for this study are supported by the safety profile of VIR-2218 in the ongoing VIR-2218-1001 (Yuen 2021) and VIR-2218-1006 studies. In VIR-2218-1001 Cohorts 1d and 1f, up to 6 doses of 200 mg VIR-2218 administered every 4 weeks either as monotherapy or in combination with PEG-IFN $\alpha$  is well tolerated and associated with deep, sustained reductions in HBsAg in patients in chronic HBV infection. In both the VIR-2218-1001 and VIR-2218-1006 studies, up to 13-dose regimens of VIR-2218 200 mg administered every 4 weeks in combination with VIR-3434 are being evaluated.



In summary, PK, safety, and antiviral activity support the VIR-2218 regimens selected for this study.

#### 4.3.3. TDF Dose Selection

TDF will be administered at a dose of 300 mg (or TD 245 mg) daily, the FDA-approved dose level and frequency for the treatment of chronic HBV infection. The optimal duration of TDF treatment is unknown and not reported in the prescribing information (VIREAD® Prescribing Information), and the patient population of the current study are not indicated for treatment. Therefore, TDF dosing will continue until the last dose of VIR-3434 and/or VIR-2218 per the respective cohort.

# 4.4. End of Study Definition

The end of study for this sub-protocol is defined as the date of the last observation of the last participant.

### 5. STUDY POPULATION

Participants that fulfil the following inclusion and exclusion criteria at screening are eligible for participation in this sub-protocol. Participants may be re-screened after consultation with the Sponsor. CCl

To achieve these characteristics, screening and/or enrollment may be restricted by the Interactive Response Technology (IRT) at any time.

## 5.1. Inclusion Criteria

# Inclusion criteria per Master Protocol, details provided for sub-protocol B in bold

- 1. Age  $\geq$  18 (or age of legal consent, whichever is older) to < 66 years
- 2. Chronic HBV infection defined as a positive serum HBsAg, HBV DNA, or HBeAg on 2 occasions at least 6 months apart based on previous or current laboratory documentation (any combination of these tests performed 6 months apart is acceptable)

In addition, as defined in Table 3 of the Master Protocol for population IV, the participants must be/have the following, within the 1-year period prior to screening:

- a. HBeAg negative
- b. HBV DNA  $\leq$  2,000 IU/mL and > LLOQ
- c. ALT ≤ ULN
- 3. Besides chronic infection with HBV, must be in good health, determined from medical history, and no clinically significant findings from physical examination, vital signs, and laboratory values
- 4. Female participants must have a negative pregnancy test or confirmation of postmenopausal status. Post-menopausal status is defined as 12 months with no menses without an alternative medical cause (see Section 10.6 for additional details). Women of child-bearing potential (WOCBP) must have a negative blood pregnancy test at screening and a negative urine pregnancy test on Day 1, cannot be breast feeding, and must be willing to use highly effective methods of contraception (Section 10.6) 14 days before study intervention administration through 48 weeks after the last dose of VIR-3434 or VIR-2218. Female participants must also agree to refrain from egg donation and in vitro fertilization from the time of study intervention administration through 48 weeks after the last dose of VIR-3434 or VIR-2218.
- 5. Male participants with female partners of child-bearing potential must agree to meet 1 of the following contraception requirements from the time of study intervention administration through 48 weeks after the last dose of VIR-3434 or VIR-2218: documentation of vasectomy or azoospermia, or male condom use plus partner use of 1 of the contraceptive options listed for contraception for WOCBP (Section 10.6). Male participants must also agree to not donate sperm from the time of first study intervention administration through 48 weeks after the last dose of VIR-3434 or VIR-2218.

6. Able to understand and comply with the study requirements and able to provide written informed consent

#### Additional Inclusion Criteria for Sub-Protocol B

- 7. HBsAg > lower limit of detection at screening
- 8. Body Mass Index (BMI)  $\geq 18 \text{ kg/m}^2 \text{ to} \leq 35 \text{ kg/m}^2$

### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

## **Exclusion Criteria per Master Protocol**

- 1. History of clinically significant liver disease from non-HBV etiology
- 2. History or current evidence of hepatic decompensation, including ascites, hepatic encephalopathy, and/or esophageal or gastric varices
- 3. History or current suspicion of malignancy diagnosed or treated within 5 years (localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screening); participants under evaluation for malignancy are not eligible.
- 4. History of bone marrow or solid organ transplant
- 5. Known active infection other than chronic HBV infection or any clinically significant acute condition such as fever (> 38° C) or acute respiratory illness within 7 days prior to Day 1
- 6. Co-infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or hepatitis E virus (HEV). Participants who are HCV antibody or HDV antibody positive, but have a documented negative HCV RNA or HDV RNA, respectively, are eligible. Participants with positive HAV immunoglobulin M (IgM) or HEV IgM but asymptomatic and with a positive HAV immunoglobulin G (IgG) or HEV IgG are eligible.
- 7. History or clinical evidence of alcohol or drug abuse within the 12 months before screening or a positive drug screen at screening unless it can be explained by a prescribed medication (the diagnosis and prescription must be approved by the investigator). Note: cannabis use is permitted
- 8. Received an investigational agent within 90 days or 5 half-lives (if known), whichever is longer, before study intervention administration or are active in the follow-up phase of another clinical study involving interventional treatment. Participants must also agree not to take part in any other interventional study at any time during their participation in this study, inclusive of the Follow-Up Period.

9. Any clinically significant medical or psychiatric condition that may interfere with study intervention, assessment, or compliance with the protocol or otherwise makes the participant unsuitable for participation in the study, as determined by the investigator.

#### Additional Exclusion Criteria for Sub-Protocol B

- 10. Significant fibrosis or cirrhosis as defined by having either a FibroScan (or sponsor-approved equivalent) result of > 8.5 kPa at screening or a liver biopsy within 1 year with Metavir F3 fibrosis or F4 cirrhosis.
- 11. History of immune complex disease
- 12. History of an autoimmune disorder
- 13. History of HBV-related extrahepatic disease, including but not limited to HBV-related rash, arthritis, or glomerulonephritis
- 14. History of allergic reactions, hypersensitivity, or intolerance to monoclonal antibodies, antibody fragments, or any excipients of VIR-3434
- 15. Prior NRTI therapy within 24 weeks prior to Day 1 or any prior therapy with PEG-IFNα
- 16. Use of any of the following systemic medications within 14 days before study intervention administration and throughout the study:
  - a. Paracetamol (acetaminophen)  $\geq 3$  g/day
  - b. Isoniazid
  - c. Systemic steroids (prednisone equivalent of > 10 mg/day) or other immunosuppressive agents (Note: corticosteroid administration for the treatment of immune-mediated AEs is allowed.)
- 17. Receipt of an oligonucleotide (eg, siRNA, antisense oligonucleotide) with activity against HBV within 48 weeks before study intervention administration
- 18. Receipt of VIR-3434 within 24 weeks prior to Day 1
- 19. Participant has the following laboratory parameters at screening by laboratory testing:
  - a. ALT > ULN at screening and any time in the 12 months prior to study enrollment
  - b. HBeAg positive at screening and any time in the 12 months prior to study enrollment
  - c. HBV DNA >2,000 IU/mL at screening and any time in the 12 months prior to study enrollment
  - d. Direct bilirubin or international normalized ratio (INR) > 1.5 ULN
- 20. Creatinine clearance (CLcr) < 30 mL/min as calculated by the Cockcroft-Gault formula at screening
- 21. Clinically significant abnormalities on 12-lead ECG at screening (as determined by the investigator)
## **5.3.** Lifestyle Considerations

Lifestyle considerations are not applicable to this study.

## **5.3.1.** Meals and Dietary Restrictions

There are no dietary restrictions in this study.

#### 5.3.2. Caffeine, Alcohol, and Tobacco

Participants that regularly consume more than 10 units of alcohol per week (1 unit = 1 glass of wine [125 mL] = 1 measure of spirits [30 mL] = one-half pint of beer [284 mL]), or more than 2 units of alcohol per day, are excluded from this sub-protocol. There are no limitations on the use of caffeine and tobacco in this study.

## 5.3.3. Activity

There are no limitations on physical activity in this sub-protocol.

#### **5.4.** Screen Failures

Participants that screen fail will not be eligible to enroll in the study. Participants may be re-screened after discussion with the Sponsor.

# 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY

# 6.1. Study Intervention(s) Administered

**Table 4:** Study Intervention (s) Administered

| Intervention Label | VIR-3434 | VIR-2218 | TDF/TD |
|---|---|---|---|
| Intervention Name | VIR-3434 | VIR-2218 | Tenofovir disoproxil<br>fumarate/ Tenofovir<br>disoproxil |
| Type | Biologic | Oligonucleotide | Drug |
| <b>Dose Formulation</b> | Lyophilized powder in vial | Liquid in vial | Tablet |
| Unit Dose<br>Strength(s) | 300 mg/vial | 200 mg/mL at 0.5mL | 300 mg tablet (TDF)<br>245mg tablet (TD) |
| Dosage Level(s) | 300 mg Q4W-Q12W | 200 mg Q4W | 300 mg QD (TDF) or<br>245 mg QD (TD) based<br>on supply source |
| Route of<br>Administration | SC | SC | Oral |
| Use | Experimental | Experimental | Experimental |
| IMP and<br>NIMP/AxMP | IMP | IMP | IMP |
| Sourcing | Sponsor | Sponsor | Sponsor |
| Packaging and<br>Labeling | Single-use vial labeled as required by country requirement. | Single-use vial labeled as required by country requirement. | Bottle labeled as required per country requirement. |
| Current or trade name(s) | VIR-3434 | VIR-2218 | Viread® |

**Table 5:** Study Arm(s)

| Arm Title | Cohort 1b | Cohort 2b |
|---|---|---|
| Arm Type | Experimental | Experimental |
| Arm Description | Participants will receive VIR-3434<br>300 mg Q4W and 300 mg TDF<br>(or TD 245 mg) QD from Day 1 to<br>Week 44 | Participants will receive VIR-3434<br>300 mg Q4W, VIR-2218 200 mg<br>Q4W and 300 mg TDF QD (or TD<br>245 mg) from Day 1 to Week 44 |
| Associated<br>Intervention Labels | VIR-3434, TDF/TD | VIR-3434, VIR-2218, TDF/TD |

## 6.2. Preparation, Handling, Storage, and Accountability

Detailed instructions for all study intervention/drugs will be provided in the Pharmacy Manual.

## 6.3. Randomization and Blinding

This is an open-label study, participants will be enrolled to one of the open cohorts in the sub-protocol.

## **6.4.** Study Intervention Compliance

Participants are expected to comply with the dosing schedule of the investigational therapies. TDF may be taken home by the participant to be administered daily per protocol. Participants will be asked to keep a treatment diary noting the day and date they take their study intervention and any adverse events. They will be asked to bring their treatment diary to each study visit along with all used and unused study intervention containers.

#### 6.5. Dose Modification

#### 6.5.1. Dose Modifications for TDF

It is recommended that TDF dose modifications be performed in accordance with the VIREAD® approved local product label.

# 6.6. Concomitant Therapy

## 6.6.1. Concomitant Therapy Not Permitted During the Study

Use of NRTIs before Day 1 is prohibited. While on the study, participants will receive TDF per protocol. No other NRTIs are permitted during the course of the Treatment Period. If participants require NRTI therapy during Follow-Up Period, Investigator may start commercial NRTI.

Use of any of the following systemic medications is prohibited within 14 days before study intervention administration and throughout the study:

- Systemic steroids (prednisone equivalent of > 10 mg/day) or other immunosuppressive agents (Note: corticosteroid administration for the treatment of immune-mediated AEs is allowed.)
- Paracetamol (acetaminophen)  $\geq 3$  g/day
- Isoniazid

Additionally, the administration of any potentially hepatotoxic medications during the study should be considered only if no therapeutic alternative can be identified and after a careful consideration of the potential risks and benefits for the participant. Medications that are potentially hepatotoxic or associated with drug-induced liver injury include, but are not limited to, the following (Björnsson 2016):

- Aspirin > 3 g/day or ibuprofen  $\ge 1.2$  g/day
- Tricyclic antidepressants
- Valproate
- Phenytoin
- Amiodarone
- Anabolic steroids
- Allopurinol
- Amoxicillin-clavulanate
- Minocycline
- Nitrofurantoin
- Sulfamethoxazole/trimethoprim
- Erythromycin
- Rifampin
- Azole antifungals
- Herbal or natural remedies

# 7. DISCONTINUATION OF STUDY, STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Study Stopping Rules

If either of the following criteria as met, dosing will be paused, and an ad hoc medical monitoring meeting will be convened with the study investigator or their representative and/or LFAC (if related to an ECI):

- 3 or more participants experience Grade 3 or higher study intervention-related AEs in the same System Organ Class (SOC)
- 2 or more participants experience Grade 4 or higher study intervention-related AEs in the same SOC

Following an assessment of all available safety data, the committee will vote to discontinue, modify (including discontinuation of one or more cohorts), or continue the study unchanged.

## 7.2. Discontinuation of Study Intervention(s)

Participants that have received at least 1 dose of VIR-3434 or VIR-2218 will not receive additional doses of either study intervention if any the following criteria are met:

- Any clinical manifestations of hepatic decompensation
- Grade 3 or higher study intervention-related AE of anaphylaxis, cytokine release syndrome, or immune complex disease
- Serum ALT  $> 10 \times ULN$
- Serum ALT or AST > 3 × ULN with any of the following laboratory results or clinical symptoms:
  - total bilirubin  $> 2 \times ULN$  or
  - INR > 1.5 × ULN (erroneously elevated INR due to incorrect blood volume collection should be ruled out) or
  - serum albumin < 3.0g/dL or
  - ascites, hepatic encephalopathy, or liver-related symptoms (eg, severe fatigue, nausea, vomiting, right upper quadrant pain in the absence of an alternative medical explanation)

The investigator should notify the medical monitor immediately in the event that any of the above criteria are met. Upon documented agreement with the investigator and the Sponsor Medical Monitor, the participant may be considered to continue receiving study intervention.

Study intervention may be discontinued in the occurrence of a condition that in the opinion of the Investigator significantly jeopardizes the wellbeing and safety of the participant. Investigator must promptly inform the Sponsor Medical Monitor if any such condition arises.

Participants who become pregnant during the Treatment Period will not receive additional doses of any study intervention. See Master Protocol for additional details.

Participants who discontinue all study interventions prematurely (eg, due to meeting a stopping rule) will undergo assessments for the EOT visit at the time of discontinuation. These participants will continue to the Follow-Up Period SOA.

# 7.3. Participant Discontinuation/Withdrawal from the Study

Refer to Master Protocol.

## 7.4. Replacement of Participants

Refer to Master Protocol.

## 7.5. Lost to Follow-up

Refer to Master Protocol.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

Study procedures and their timing are summarized in SOA (Section 10.9). Refer to Master Protocol for additional details

## 8.1. Screening Period

Refer to Master Protocol.

## 8.2. Efficacy Assessments

Refer to Master Protocol.

## 8.3. Safety Assessments

Planned timepoints for all safety assessments are provided in the SOA.

#### **8.3.1.** Physical Examinations

Refer to Master Protocol. In addition to the Master Protocol:

- At screening, body weight and height will be measured, and BMI will be calculated.
- Body weight will also be measured at study visits as indicated in the SOA.

## 8.3.2. Vital Signs

Refer to Master Protocol.

#### **8.3.3.** Clinical Safety Laboratory Tests

Clinical laboratory tests that will be performed in this study are presented in Section 0. In the event of an unexplained clinically relevant (in the opinion of the investigator) abnormal laboratory test occurring after study intervention administration, the test may be repeated and followed up at the discretion of the investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

### 8.3.4. Pregnancy Testing

Please refer to Master Protocol.

### 8.3.5. Local Tolerability

If a local reaction around the injection site occurs, photographs may be obtained. Participants should be instructed to monitor for local and systemic ISRs, including signs and symptoms of anaphylaxis and instructed to seek emergency medical care, if needed. Oral analgesics may be used to manage mild to moderate local pain or tenderness. More extensive or severe symptoms (eg, suspected anaphylaxis, cytokine release syndrome, or immune complex disease) should be evaluated by the study investigator and treated as deemed appropriate by the investigator and per local standards of care. See Section 10.8 for additional details.

# 8.4. Assessment of Viral Parameters, Antiviral Activity, and Resistance Surveillance

In addition to Master Protocol, assessments of antiviral activity performed after screening will include: HBsAg (quantitative), anti-HBs (quantitative), HBeAg (qualitative or quantitative as specified in the SOA), anti-HBe, and HBV DNA.

Assessments of exploratory viral markers or other viral analyses may also be performed after screening as described in the Master Protocol.

Resistance surveillance to monitor for the potential development of resistance to NRTI (TDF), VIR-3434, or VIR-2218 will be conducted for all participants who receive study intervention. HBV genome sequencing will be attempted in participants with HBV DNA rebound as defined by HBV DNA  $\geq 500$  IU/mL. As it will not be known at the time of visit if a participant has virologic rebound, samples for resistance surveillance will be collected at all study visits noted in the SOA. Samples collected for resistance surveillance may be used to perform additional viral analyses, including but not limited to viral sequencing.

Details regarding the processing and shipping of the samples are provided in the Laboratory Manual.

## 8.5. **CCI**

CCI Time points for assessments are provided in the SOA for each applicable cohort.

# **8.6.** Exploratory Assessments

#### **8.6.1.** Exploratory Analysis Samples

Refer to Master Protocol.

## 8.6.2. **CCI**

Details regarding the processing, shipping, and analysis of these samples are provided in the Laboratory Manual.

### 8.6.2.1. **CCI**

Refer to Master Protocol.

### 8.6.2.2. **CCI**

Refer to Master Protocol.

#### 8.6.2.3. **CCI**

Refer to Master Protocol.

#### 8.6.3. **CCI**

#### CCI

Samples

will be collected at certain time points per the SOA for a given cohort. Details regarding sample processing, shipping, and storage are provided in the Laboratory Manual and Vir Immunology Sample Manual (if applicable).

## CCI

Based on emerging data, the Sponsor may restrict enrollment to certain sites or cohorts.

# 8.7. Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Safety Reporting

Refer to Master Protocol.

#### 8.7.1. Time Period and Frequency for Collecting AE and SAE Information

Refer to Master Protocol.

#### 8.7.2. Follow-up of AEs and SAEs

Refer to Master Protocol.

## 8.7.3. Regulatory Reporting Requirements for SAEs

Refer to Master Protocol.

#### 8.7.4. Adverse Events of Interest

Not applicable

# 8.7.5. Clinical Laboratory Abnormalities and Other Abnormal Assessments as AEs or SAEs

Refer to Master Protocol.

## 8.7.6. Laboratory Events of Clinical Interest

Laboratory ECI for this study are defined as instances of ALT > 3x ULN.

An ECI is considered resolved when ALT returns to  $\leq$  ULN.

All ECIs must be reported to the Sponsor Medical Monitor within 5 business days of the investigator becoming aware of the ECI. In addition, the assessments outlined in Section 10.7 should be performed as soon as possible and no later than two weeks after the initial ALT value meeting criteria for a laboratory ECI.

## 8.7.7. Special Situation Reports

Refer to Master Protocol.

## **8.7.7.1. Pregnancy**

Refer to Master Protocol.

#### 8.8. Pharmacokinetic Assessments

Blood samples will be collected to assess concentrations of VIR-3434 and VIR-2218 (for cohorts receiving VIR-2218). Timepoints for the collection of samples for VIR-3434 and VIR-2218 PK analysis are provided in the SOA. Concentrations of VIR-3434 and VIR-2218 PK will be quantified using a validated bioanalytical assay. These assessments are exploratory and may or may not be analyzed. Specific assays used for these assessments may be changed at the Sponsor's discretion based on emerging data. Details regarding the processing, shipping, and analysis of the samples are provided in the Laboratory Manual.

# 8.9. Immunogenicity Assessments

Blood samples will be collected for analysis of immunogenic responses to determine presence/absence and titers of ADA as applicable, according to the timepoints defined in the SOA. Samples may also be characterized for neutralizing potential of anti-VIR-3434 antibody (NAb), as appropriate. Details regarding the processing, shipping, and analysis of the samples are provided in the Laboratory Manual.

## 8.10. Electrocardiogram

12-lead safety ECGs will be recorded and reviewed on-site by the investigator. ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. All ECGs should be measured in the supine position after the participant has rested comfortably for approximately 10 minutes. ECG should be measured before blood sample collection and administration of study intervention(s), where applicable.

## 8.11. Liver Elastography (eg, FibroScan)

To exclude the presence of cirrhosis, participants will have a liver elastography (eg, FibroScan or other sponsor-approved method) evaluation. This is not required to be performed if the participant has had a liver elastography in the 6 months prior to screening or liver biopsy in the year prior to screening that confirmed the absence of Metavir F3 fibrosis or F4 cirrhosis.

### 9. STATISTICAL CONSIDERATIONS

This section provides a summary of the planned statistical analyses. Details of the statistical analyses will be provided in the Statistical Analysis Plan (SAP), which will be finalized prior to first interim analysis and database lock.

Any change to the data analysis methods described in the protocol will require an amendment only if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol and the justification for making the change will be described in the SAP and/or the clinical study report. Additional exploratory analyses of the data will be conducted as deemed appropriate.

## 9.1. Statistical Hypotheses

The null hypothesis is that the response rate, defined as the proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) at EOT, is  $\le$  2%, which is the assumed rate of HBsAg loss in NRTI-suppressed patients. The alternative hypothesis is that the response rate is greater than 2%.

This study is exploratory in nature. No multiplicity adjustment will be made.

## 9.2. Sample Size Determination

A sample of 15 in each cohort will provide approximately 76% statistical power for each cohort to reject the null hypothesis, if the true HBsAg loss rate is 25%, using a 1-sided exact binomial test with a significance level of 2.5%.

Up to 30 participants will be enrolled in this sub-protocol initially. Additionally, up to 30 floater participants may be added to the cohorts at any time at Sponsor's discretion. As described in Section 9.5, this addition may be based on the data from interim analysis. No more than 60 participants will be enrolled.

## 9.3. Analysis Sets

In addition to the Master Protocol, the following analysis sets will apply to this sub-protocol:

| Analysis Sets | Description |
|---|---|
| PK Analysis Set | The PK Analysis Set includes all participants in the Full Analysis Set who had at least one measurable postdose concentration. |
| | The PK Analysis Set will be used for all PK analyses. |
| Immunogenicity Analysis Set | Immunogenicity Analysis Set includes all participants in the Full Analysis Set who had at least 1 postdose measurement of immunogenicity, including screening, titer, or neutralizing characterization, as applicable |
| | The Immunogenicity Analysis Set will be used for analyses of the immunogenicity endpoints. |
| | Details of immunogenicity analyses will be provided in the SAP. |

## 9.4. Statistical Analyses

#### 9.4.1. General Considerations

Refer to the Master Protocol.

TEAE definition for this sub-protocol: An AE that is reported with an onset date on or after the start of study intervention(s) until end of Follow-Up Period.

Prior to the final analysis, interim analyses will be conducted, and the analyses may be submitted for publication or to regulatory agencies to seek guidance for the overall clinical development program.

## 9.4.2. Primary Endpoint(s) Analysis

The primary efficacy endpoint is the proportion of participants achieving suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) at EOT.

#### 9.4.2.1. Target Population

All eligible participants with chronic HBV infection, as defined in the Full Analysis Set.

#### 9.4.2.2. Population Level Summary

The proportion of participants who achieved suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) at EOT and the corresponding two-sided 95% exact Clopper-Pearson confidence intervals.

## 9.4.3. Secondary Endpoint(s) Analysis

Refer to the Master Protocol for the safety data analysis.

The key secondary efficacy endpoints (see Section 3 in this protocol and the PREVAIL Master Protocol) including the effect of the study intervention on HBsAg, anti-HBs, HBeAg, and HBV DNA in the Full Analysis Set will be summarized.

#### 9.4.4. Exploratory Endpoint(s) Analysis



Missing data due to withdrawal or all other events will not be imputed.

## 9.4.5. Missing Data

Values for missing safety laboratory data will not be imputed. However, a missing baseline result (defined as predose Day 1) will be replaced with a screening result, if available.

If no pre-treatment laboratory value is available, the baseline value will be assumed to be normal (ie, no grade [Grade 0]) for the summary of graded laboratory abnormalities. If safety laboratory results for a participant are missing for any reason at a time point, the participant will be excluded from the calculation of summary statistics for that time point.

## 9.4.6. Other Safety Analyses

Refer to the Master Protocol for other safety data analysis.

## 9.5. Interim Analysis





## 9.6. Pharmacokinetic Analyses

VIR-2218 and VIR-3434 concentration data from all sparse samples may be pooled with data from other studies and may be used for estimation of population PK parameters.

PK/pharmacodynamic analyses will be conducted to explore exposure-response relationships between PK parameters and selected antiviral variables. These analyses may include graphical plots, tabular summaries, and various linear and/or nonlinear analyses. Details of the analysis will be provided in a separate analysis plan.

# 9.7. Immunogenicity Analyses

For all study parts, immunogenicity data will be listed and summarized using descriptive statistics, including incidence, titers, and neutralization data, as applicable.

Correlations between immunogenicity data and safety, efficacy, and PK data will be explored. These analyses may include graphical plots, tabular summaries, and various linear and/or nonlinear analyses. Details of immunogenicity analyses will be provided in the SAP.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

#### 10.1.1. Regulatory and Ethical Considerations

Refer to Master Protocol.

#### 10.1.2. Financial Disclosure

Refer to Master Protocol.

#### 10.1.3. Informed Consent Process

Refer to Master Protocol.

#### 10.1.4. Data Protection

Refer to Master Protocol.

#### 10.1.5. Confidentiality

Refer to Master Protocol.

#### 10.1.6. Committees Structure

### 10.1.6.1. Liver Flare Adjudication Committee (LFAC)

The LFAC will provide hepatic safety oversight by performing periodic reviews of data pertaining to participants who meet certain prespecified criteria for transaminase elevations Section 8.7.6. Additionally, the Sponsor may request LFAC evaluation of specific patient data at any time. The LFAC will be governed by an LFAC Charter that will be finalized prior to screening the first participant. The LFAC membership composition, laboratory criteria to trigger patient case evaluation by the LFAC, and data review requirements are described in detail in the LFAC Charter.

#### 10.1.7. Dissemination of Clinical Study Data

Refer to Master Protocol.

#### **10.1.8.** Data Quality Assurance

Refer to Master Protocol.

#### **10.1.9. Source Documents**

Refer to Master Protocol.

#### 10.1.10. Electronic Case Report Forms (eCRF)

Refer to Master Protocol.

## 10.1.11. Study and Site Start and Closure

Refer to Master Protocol.

## 10.1.12. Publication Policy

Refer to Master Protocol.

# **10.2.** Appendix 2: Clinical Laboratory Tests

**Table 6:** Protocol-Required Safety Laboratory Tests

| Chemistry | Hematology |
|---|---|
| Albumin Blood urea nitrogen (BUN) Calcium Bicarbonate Chloride Creatine kinase <sup>a</sup> Creatinine Creatinine clearance (calculated) <sup>b</sup> Gammaglutamyltransferase (GGT) Glucose (non-fasting) Lactate dehydrogenase (LDH) Phosphate Potassium Sodium Liver Function Tests: Alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (total and direct) Complement (C3, C4, CH50) <sup>c</sup> | Platelet count Red blood cell (RBC) count Hemoglobin Hematocrit White blood cell (WBC) count with differential: neutrophils, lymphocytes, monocytes, eosinophils, basophils RBC indices: mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), % reticulocytes |
| Coagulation Parameters | Pregnancy Testing |
| International normalized ratio (INR) Prothrombin time (PT) | Highly sensitive (serum/plasma or urine) human chorionic gonadotropin (hCG) pregnancy test (as needed for women of childbearing potential) |

| Urinalysis | Additional Screening Tests |
|---|---|
| Bilirubin Glucose Ketones Leukocytes Microscopy (if blood or protein is abnormal) Nitrite pH Proteins RBCs Specific gravity Urobilinogen Visual inspection for appearance and color | Urine drug screen (to include at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines) Serology: Hepatitis A <sup>d</sup> , B, C <sup>e</sup> , D <sup>f</sup> and E <sup>d</sup> Human immunodeficiency virus I and II Lipase Amylase Follicle stimulating hormone (FSH) <sup>g</sup> Hemoglobin A1c (HbA1c) Thyroid stimulating hormone (TSH) Free T4 HBV genotyping |

<sup>&</sup>lt;sup>a</sup> Only required if ALT and/or AST is elevated > 2x the predose Day 1 baseline value

<sup>&</sup>lt;sup>b</sup> Please note the following clarification for the creatinine clearance calculation: for study visits where weight is not measured, creatinine clearance will be calculated using the value measured from the most recent study visit.

<sup>&</sup>lt;sup>c</sup> As indicated in the Schedule of Activities (Section 10.9)

<sup>&</sup>lt;sup>d</sup> Participants with positive HAV IgM or HEV IgM but asymptomatic and with a positive HAV IgG or HEV IgG are eligible.

<sup>&</sup>lt;sup>e</sup> Participants with positive HCV screening serology may have HCV RT-PCR performed to determine eligibility.

<sup>&</sup>lt;sup>f</sup> Participants with positive HDV screening serology may have HDV RNA performed to determine eligibility.

<sup>&</sup>lt;sup>g</sup> Required for confirmation of menopause only as applicable

# 10.3. Appendix 3: AEs, SAEs, SSRs and AEIs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

Refer to Master Protocol.

## 10.4. Appendix 4: List Abbreviations and Definitions of Terms

ADA anti-drug antibodies

ADCC/ADCP antibody dependent cellular toxicity/antibody dependent cellular

phagocytosis

ALP alkaline phosphatase
ALT alanine aminotransferase
AST aspartate aminotransferase

BMI body mass index
BUN blood urea nitrogen
DNA deoxyribonucleic acid
ECG electrocardiogram

ECI events of clinical interest

EOT end of treatment

#### CCI

FcRn Fc receptor

FSH follicle stimulating hormone
GGT gammaglutamyltransferase

HAV hepatitis A virus

HBcrAg hepatitis B correlated antigen

HBeAg hepatitis B e antigen

HBIG hepatitis B immune globulin

HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma

HCV hepatitis C virus
HDV hepatitis D virus
HEV hepatitis E virus

HIV human immunodeficiency virus

IB Investigator's Brochure
IgG immunoglobulin G
IgM immunoglobulin M

INR international normalized ratio
IRR infusion related reaction

IRT Interactive Response Technology

ISR injection site reaction

LDH lactate dehydrogenase

LFAC Liver Flare Adjudication Committee

mAb monoclonal antibody

MCH mean corpuscular hemoglobin
MCV mean corpuscular volume
NAb neutralizing antibodies

NRTI nucleos(t)ide reverse transcriptase inhibitors

NSAID non-steroidal anti-inflammatory drug
PBMC peripheral blood mononuclear cells

PEG-IFNα peginterferon-alfa-2a
PK pharmacokinetics
PT prothrombin time

QD once a day
Q4W every 4 weeks
Q12W every 12 weeks
RBC red blood cell

SAP Statistical Analysis Plan

siRNA small interfering ribonucleic acid

SOA Schedule of Activities

SRC safety review committee

TD tenofovir disoproxil

TDF tenofovir disoproxil fumarate

TND target not detected

TSH thyroid stimulating hormone

ULN upper limit of normal

WBC white blood cell

WOCBP women of child-bearing potential

# 10.5. Appendix 5: Summaries of Changes for Previous Protocol Amendments

## Protocol Amendment 2 (11 October 2022) Summary of Changes Table

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| <ul><li>1.1 Synopsis</li><li>3. Objectives and Endpoints</li><li>9. Statistical Considerations</li></ul> | Added assessment of hepatitis B virus (HBV) DNA suppression (< lower limit of quantitation [LLOQ]) at the end of treatment to the primary endpoint Added proportion of participants achieving hepatitis B surface antigen (HBsAg loss (< 0.05 IU/mL) at the end of treatment to the secondary endpoints. | The prior primary endpoint to evaluate proportion of participants achieving HBsAg loss (<0.05 IU/mL) at the end of treatment was moved to be a secondary endpoint and the primary endpoint was modified to include HBV DNA suppression ( <lloq) (<0.05="" (fda="" 2022).<="" align="" and="" at="" better="" both="" clinical="" effect="" end="" fda="" for="" guidance="" hbsag="" hbv="" interventions="" iu="" loss="" ml)="" of="" on="" parameters="" study="" td="" the="" treatment="" understanding="" viral="" with=""></lloq)> |
| 1.1. Synopsis 1.2. Study Schema 3. Objectives and Endpoints 4.1.2.1. Intervention Groups 4.1.2.3.2. Treatment Period 4.2.1. Rationale for VIR-3434 for the Treatment of Chronic HBV Infection 4.2.3. Rationale for VIR-3434 + VIR-2218 + TDF for the Treatment of Chronic HBV Infection 6.1. Study Intervention(s) Administered 9.4.1. General Considerations 10.9. Appendix 9: Schedule of Activities | Removed option for participants to discontinue study intervention at Week 20 and move into the Follow-up Period if they achieve undetectable HBsAg and HBV DNA < LLOQ at 2 consecutive visits by Week 20. As a result of this change, dosing of study intervention and duration of treatment was updated for Cohorts 1b and 2b, and the exploratory endpoint assessing proportion of participants with HBsAg loss maintained 24 weeks post-end of treatment (EOT) of Week 20 was removed. | Removal of the option to discontinue treatment early would allow for all participants within the cohort to receive the same duration of treatment and thereby allow consistency of analyses of the regimen. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 2.3.1. Risk Assessment | Updated immunogenicity risks for VIR-2218 and VIR-3434. Additional edits were made to terminology and definitions to align with the most recent VIR-2218 and VIR-3434 Investigator's Brochures (IBs). | To provide updated risk assessment information for VIR-2218 and VIR-3434 per the most recent IBs. |
| 4.1.3. NRTI Treatment | Added additional criteria for which commercial nucleos(t)ide reverse transcriptase inhibitors (NRTI) therapy be initiated in participants at any time during the Follow-up Period | Additional criteria were added to ensure prompt identification of participants that may be at a risk for safety complications. Recommendation for treatment with NRTI and additional safety monitoring for these participants are outlined in Section 4.1.3. |
| <ul><li>5.2. Exclusion Criteria</li><li>8.11. Liver Elastography (new section)</li><li>10.9. Appendix 9: Schedule of Activities</li></ul> | Clarified that, in addition to FibroScan, liver elastography can be assessed with other Sponsorapproved methods | Some study sites may not have access to FibroScan to measure liver elastography. Sponsor may approve alternate methods to determine fibrosis in these cases. |
| 5.2. Exclusion Criteria 8.10. Electrocardiogram 10.9. Appendix 9: Schedule of Activities | Added Exclusion Criterion #21: Clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening (as determined by the investigator) In addition to at screening, added 12-lead safety ECGs assessments at Day 8 in the Treatment Period and Follow-up Period. | Screening and post-dose safety ECG assessments have been added to assess cardiac safety. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 7.1. Study Stopping Rules | Added study stopping rules | Criteria were added to trigger an ad hoc medical monitoring meeting in which a recommendation to discontinue, modify, or continue the study will be made. |
| 8.3.1. Physical Examinations 10.9. Appendix 9: Schedule of Activities | In addition to at screening, body weight measurements were also added at study visits as indicated in the Schedule of Activities. | Body weight is required to calculate creatinine clearance. |
| 9.3. Analysis Sets | Modified pharmacokinetic (PK) Analysis Set to include all participants in the Full Analysis Set (previously All Enrolled Set) who received at least one dose of study drug and had at least one measurable postdose concentration. Modified Immunogenicity Analysis Set to include all participants in the Full Analysis Set (previously Safety Analysis Set) who had at least one postdose measurement of immunogenicity. | To align with the updated definition of the Full Analysis Set in the master protocol. The Full Analysis Set includes all participants who received at least one dose of study intervention(s) irrespective of post-dose assessments. |
| 9.6. Pharmacokinetic Analyses | Clarified that VIR-2218 and VIR-3434 concentration data from all sparse PK samples may be pooled with data from future studies and may be used for estimation of population PK parameters. | To provide updated PK analyses plan |
| 10.6. Appendix 6: Contraceptive and Barrier Guidance | Clarified that an elevated follicle stimulating hormone (FSH) in the post-menopausal range should be used to confirm a post-menopausal state in women not using hormonal contraception or hormone replacement therapy. | To correct FSH criteria used to confirm a post-menopausal state. |
| 10.9. Appendix 9: Schedule of Activities | Added additional visits in the Follow-up Period at Weeks 2, 6, 10, 28, 32, 40, and 44. | More frequent visits after completion of treatment period were added to ensure prompt identification of any participants that may be at a risk for safety complications. |
| Entire document | Other administrative, formatting, and other minor changes | These changes were made to clarify, ensure consistency, provide up-to-date information, or rectify typographical errors. |

## Protocol Amendment 1 (16 May 2022) Summary of Changes Table

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Study title | Modified study title to "A Phase 2 Study Evaluating the Efficacy and Safety of VIR-3434 and/or VIR-2218 containing regimens in HBeAg-negative Participants with Low Viral Burden of Chronic Hepatitis B Infection (THRIVE)" | Study title was modified to be concise |
| 1.1 Synopsis 3. Objectives, endpoints and estimands 9.4.2 Primary Endpoint Analysis | Moved one co-primary endpoint (Proportion of participants with HBsAg loss at 24 weeks postend of treatment) to be a secondary endpoint, making "Proportion of participants with HBsAg loss (< 0.05 IU/mL) at the end of treatment" the only primary endpoint | This modification was made to focus the primary endpoint of the study to understand the proportion of participants that achieve HBsAg loss on-treatment. The sustained HBsAg loss and any additional off-treatment HBsAg loss will be evaluated as secondary endpoints in this study. |
| 1.1 Synopsis 3. Objectives, endpoints and estimands | Added secondary endpoints #10 and 14 and modified #11 # 10 Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) after discontinuation of all treatment at 24 weeks at 48 weeks #11 Proportion of participants achieving sustained suppression of HBV DNA (< LLOQ) with HBsAg loss (< 0.05 IU/mL) after discontinuation of all treatment at 24 weeks at 48 weeks at 48 weeks | Endpoints 10, and 11 were added/modified to conform with the FDA HBV clinical guidance (FDA 2022). Endpoint 14 was added for better understanding of the change in HBsAg levels through the study. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.1 Synopsis 3. Objectives, endpoints and estimands | <ul> <li>Moved these secondary endpoints and the respective objectives to exploratory endpoints</li> <li>Proportion of participants meeting criteria for NRTI treatment in Follow-Up Period</li> <li>HBV DNA levels and change from baseline across timepoints in the study</li> <li>Nadir and maximum change of HBV DNA levels from baseline in the study</li> </ul> | These endpoints will provide additional understanding of the changes in the HBV DNA and of participants needing NRTI treatment after end of treatment. Therefore, they were better suited as exploratory endpoints |
| 1.1 Synopsis 3. Objectives, endpoints and estimands | Added exploratory objective and corresponding endpoint #11 Proportion of participants with virological relapse (defined as either (1) an increase of $\geq 1 \log 10 \ HBV \ DNA \ IU/mL$ above nadir for at least 2 consecutive visits $OR$ (2) quantifiable $HBV \ DNA \ of \geq 1 \log 10 \ IU/mL$ above $LLOQ$ for at least 2 consecutive visits after being $\langle LLOQ \rangle$ | This endpoint was added to conform to the FDA HBV clinical guidance to evaluate any virological relapse. This will distinguish virological relapse from transient increases in HBV DNA that are possible after discontinuing NRTI (FDA 2022). |
| 1.1 Synopsis 3. Objectives, endpoints and estimands | Other minor clarifications to primary and secondary endpoints: Defining HBsAg loss as < 0.05 IU/mL Modifying TND or undetectable HBV DNA across different secondary endpoints as < LLOQ | These changes were made to provide clarifications to the level of viral marker referenced. The HBV DNA level was modified from being TND (target not detected) to < LLOQ to conform to the FDA guidance (FDA 2022) |
| 4.1 Overall study design<br>Table | Participant population including in this sub-<br>protocol was modified from HBV DNA<br>< 2,000 IU/mL and ALT < ULN to be HBV DNA<br>≤ 2,000 IU/mL and ALT ≤ ULN | This modification was made to include participants that may have the limit values and to align with major clinical practice guidelines (Terrault 2018 and EASL 2017) |
| 4.1.2.3.2 Treatment Period | Criteria to stop study interventions at W20 for Cohorts 1b and 2b were modified to include HBV DNA < LLOQ in addition to undetectable HBsAg | This criterion was added to ensure that participants that stop study interventions have achieved HBV DNA suppression and thereby increasing the probability of long-term sustained suppression off-treatment. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 4.1.2.3.4 NRTI treatment during Follow-Up | Added criteria to consider starting NRTI in the Follow-Up Period if "any other clinically significant event(s) warranting the NRTI therapy in the opinion of the investigator occur". | This criterion was added to ensure investigator had the option to start NRTI treatment with any clinical event(s) that in their opinion may affect participant safety after discontinuation of all study treatments. |
| 5.2 Exclusion criteria | Exclusion criterion #23 from "Prior NRTI therapy" to "Prior NRTI therapy within 24 weeks prior to Day 1 or any prior therapy with PEG-IFNa" | This criterion was modified to allow inclusion of participants that may have had prior NRTI therapy but have been off NRTIs for at least 24 weeks prior to dosing in the current study. Prior PEG-IFNα was added as an exclusion to allow assessment of participants that were not PEG-IFNα-experienced and provide a clear understanding of the safety and efficacy of the current study regimens |
| 9.3 Analysis Sets | Clarified that the PK and immunogenicity analysis sets will include all participants from the Safety Analysis Set who received at least one dose of study drug and had at least one measurable post-dose concentration or at least one post-dose immunogenicity measurement respectively. | Modified to provide clarity |
| Entire document | Other administrative, formatting, and other minor changes | These changes were made to clarify, ensure consistency, or rectify typographical errors. |

## 10.6. Appendix 6: Contraceptive and Barrier Guidance

WOCBP may be included in this study and include any female participant who has experienced menarche and who is not post-menopausal or permanently sterilized (eg, bilateral tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

 WOCBP must be willing to use highly effective methods of contraception from 14 days before the first dose of study intervention to 48 weeks after the final dose of VIR-3434 or VIR-2218. After the end of study, use of TDF in WOCBP should be determined per the VIREAD® approved local product label.

Highly effective methods of birth control are defined as those that result in a low failure rate (ie, less than 1% per year). Birth control methods which are considered highly effective include:

- Established use of combined (estrogen and progestogen containing) oral, intravaginal, or transdermal hormonal methods of contraception associated with inhibition of ovulation OR established use of progestogen-only oral, injectable, or implantable hormonal methods of contraception associated with inhibition of ovulation. It is not currently known whether VIR-2218 or VIR-3434 will impact the effectiveness of hormonal contraceptive methods; therefore, it is recommended to use an additional form of contraception (ie, barrier method) for 48 weeks after the last administration of VIR-3434 or VIR-2218. After the end of study, use of TDF in WOCBP should be determined per the VIREAD® approved local product label.
- Placement of an intrauterine device
- Placement of an intrauterine hormone-releasing system
- Surgical sterilization of male partner (with the appropriate documentation of vasectomy or the absence of sperm in the ejaculate; for female participants on the study, the vasectomized male partner should be the sole partner for that participant)
- True sexual abstinence from heterosexual contact, when in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent participants must agree to use 1 of the above-mentioned contraceptive methods for 48 weeks after last dose of VIR-3434 or VIR-2218 if they start heterosexual relationships during the study. After the end of study, use of TDF in WOCBP should be determined per the VIREAD® approved local product label.
- Barrier method in combination with hormonal contraceptive, as described above

Post-menopausal status is defined as 12 months with no menses without an alternative medical cause. An elevated follicle stimulating hormone (FSH) level in the post-menopausal range should be used to confirm a post-menopausal state in women not using hormonal contraception or hormone replacement therapy (HRT). In the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.

Females on HRT and whose menopausal status is in doubt must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

Female participants must also agree to refrain from egg donation and in vitro fertilization from the time of study intervention administration through 48 weeks after the last dose of VIR-3434 or VIR-2218. After the end of study, use of TDF in WOCBP should be determined per the VIREAD® approved local product label.

Male participants with female partners of child-bearing potential must agree to meet 1 of the following contraception requirements from the time of study treatment administration until 48 weeks after the last administration of VIR-3434 or VIR-2218. After the end of study, use of TDF in males with female partners of child-bearing potential should be determined per the VIREAD® approved local product label.

- Documentation of azoospermia or vasectomy
- Male condom plus partner use of 1 of the contraceptive options listed above for contraception for WOCBP (hormonal contraceptive, intrauterine device)

Male participants must also agree not to donate sperm from the first dose of study intervention through 48 weeks after the last dose of VIR-3434 or VIR-2218. After the end of study, use of TDF in males donating sperm should be determined per the VIREAD® approved local product label.

# 10.7. Appendix 7: Additional Assessments in Participants That Experience ALT Elevation Meeting ECI Criteria

Additional assessments will be performed in participants who experience ALT elevations meeting ECI criteria as outlined in Section 8.7.6. Following the occurrence of elevated ALT meeting ECI criteria per central laboratory, the assessments in Table 7 will be performed as soon as possible and no later than 2 weeks after the initial ALT value meeting criteria for a laboratory ECI.

The full panel of assessments should only be performed once per ECI occurrence. An ECI occurrence is considered resolved when ALT returns to  $\leq$  ULN.

Individual assessments may be repeated per investigator discretion, as needed.

Participants who meet ECI criteria will continue to receive study intervention unless criteria for study intervention discontinuation are met. Criteria for individual patient discontinuation from further dosing are described in Section 7.1.

Table 7: Assessments in Participants That Experience ALT Elevation Meeting ECI Criteria

| Chemistry | Hematology |
|---|---|
| Albumin Blood urea nitrogen (BUN) Calcium Bicarbonate Chloride Calcium Creatine kinase Creatinine Creatinine clearance (calculated) Gammaglutamyltransferase (GGT) Glucose Lactate dehydrogenase (LDH) Phosphate Potassium Sodium Uric acid Lipase Liver Function Tests: Alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (total and | Platelet count Red blood cell (RBC) count Hemoglobin Hematocrit White blood cell (WBC) count with differential: neutrophils, lymphocytes, monocytes, eosinophils, basophils RBC indices: mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), % reticulocytes |
| direct) Coagulation Parameters | Exploratory testing |
| International normalized ratio (INR) Prothrombin time (PT) | CCI CCI CCI CCI |

| Extended Hepatic Panel | Imaging |
|---|---|
| Quantitative HBsAg | Abdominal ultrasound, including doppler flow if |
| HBV DNA | available (CT or MRI is acceptable in place of |
| Quantitative HBeAg | ultrasound if clinically indicated) |
| HAV antibody IGM | |
| HCV antibody | |
| HCV RNA PCR (qualitative and quantitative) | |
| HDV antibody or RNA | |
| HEV antibody IgM | |
| Epstein-Barr Virus antibodies (IgM and IgG) Cytomegalovirus antibodies (IgM and IgG) | |
| Varicella Zoster Virus antibodies IgG | |
| HSV-I and II IgG | |
| IgG | |
| Phosphatidylethanol | |
| Aldolase | |
| Anti-nuclear antibodies Anti-Smooth muscle antibodies | |
| Anti-LKM1 antibody | |
| Anti-nitochondrial antibodies | |
| Anti-SLA antibodies | |
| Ferritin | |
| Ceruloplasmin | |
| IgM | |
| Urinary ethylglucuronide | |
| Acetaminophen | |
| <b>Focused Medical History</b> | |
| Use of any potentially hepatotoxic concomitant medications, including over the counter medications and herbal remedies | |
| Exposure to other potentially hepatotoxic agents including any work-related exposures (eg, solvents, pesticides, etc.) | |
| Alcohol consumption and drugs of abuse | |
| Travel history | |
| Exercise History | |

# 10.8. Appendix 8: Anaphylaxis, Cytokine Release Syndrome, And Immune Complex Disease Supportive Measures

The following equipment or agents may be needed in the event of a suspected anaphylactic reaction or cytokine release syndrome:

- ECG monitor
- Blood pressure monitor
- Oxygen saturation monitor
- Thermometer
- Tourniquet
- Oxygen
- Mechanical ventilator
- Renal replacement therapy
- IV infusion solutions, tubing, catheters, and tape
- Fresh-frozen plasma and/or cryoprecipitate
- Epinephrine
- Antihistamines, such as diphenhydramine
- Corticosteroids, such as hydrocortisone, prednisolone, and methylprednisolone

The following are procedures that may be followed in the event of a suspected anaphylactic reaction or cytokine release syndrome:

- Maintain an adequate airway
- Stop study intervention injection (if reaction occurs during injection)
- Call for additional medical assistance
- Apply a tourniquet proximal to the injection site to slow systemic absorption of study intervention (if reaction occurs during injection). Do not obstruct arterial flow in the limb.
- Ensure appropriate monitoring is in place, such as continuous ECG and pulse oximetry monitoring
- Administer epinephrine, antihistamines, corticosteroids or other medications/products as necessary based on the status of the participant and as directed by the physician
- Draw local laboratory samples as appropriate, possibly including evaluation of cytokines
- The following equipment or agents may be needed in the event of suspected immune complex disease
- Thermometer

- Analgesic and antipyretic agents, such as non-steroidal anti-inflammatory drugs (NSAIDs)
- Antihistamines, such as diphenhydramine
- Corticosteroids, such as prednisone and methylprednisolone
- In extreme cases, equipment for plasmapheresis may be needed

The following are procedures that may be followed in the event of suspected immune complex disease:

- Though unlikely to occur acutely, stop study intervention injection (if reaction occurs during injection)
- Ensure temperature is appropriately monitored
- Monitor for most common manifestations, including rheumatic (arthralgias) and dermatologic (pruritic rash) findings
- Administer NSAIDs, antihistamines, corticosteroids, or other medications/products as necessary based on the status of the participant and as directed by the physician
- Draw local laboratory samples as appropriate, possibly including complete blood count, erythrocyte sedimentation rate, C-reactive protein, urinalysis, serum chemistry, and evaluation of complement
- In extreme cases, plasmapheresis may be employed

# 10.9. Appendix 9: Schedule of Activities

Assessments in **bold** are in addition to those listed in the PREVAIL Master Protocol.

**Table 8:** Schedule of Activities: Cohort 1b

| Study Stage | Screening | Treatment Period <sup>a</sup> | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | , | V1 | W4 | W8 | W8 W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to D-1 | D1 | D8 ±2 | D29±2 | D57±2 | D85±2 | D113±2 | D141±2 | D169±2 | D197±2 | D225±2 | D253±2 | D281±2 | |
| Study Procedures | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | Xc | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | |
| Physical examination | X | | | | | | | | | | | | | X |
| Body Weight | | | | | | | X | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Vital signs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse event review/record <sup>e</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Liver elastography (eg, Fibroscan) f | X | | | | | | | | | | | | | |
| 12-lead safety ECG <sup>g</sup> | X | | X | | | | | | | | | | | |
| ECI surveillanceh | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| VIR-3434 local tolerability i | | X | | | | | | | | | | | | |
| Drug Administration | | - | • | | | | • | | | | | | | |
| VIR-3434 administration <sup>j</sup> | | X | | X | X | X | X | X | X | X | X | X | X | X |
| TDF administration (QD) k | | | • | | | | • | X | • | • | | | | |

| Study Stage | Screening | Treatment Period <sup>a</sup> | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | W1 | | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to D-1 | D1 | D8 ±2 | D29±2 | D57±2 | D85±2 | D113±2 | D141±2 | D169±2 | D197±2 | D225±2 | D253±2 | D281±2 | |
| CCI | , | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | |
| Treatment Diary | | | | | | | | X | | | | | | |
| Laboratory Assessments <sup>m</sup> | | | | | | | | | | | | | | |
| Pregnancy test <sup>n</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Screening viral serology o | X | | | | | | | | | | | | | |
| Liver function tests <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum chemistry <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation parameters <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis <sup>pq</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine for drugs of abuse r | X | | | | | | | | | | | | | |
| HBsAg quantitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Anti-HBs qualitative | X | | | | | | | | | | | | | |
| Anti-HBs quantitative | | X | | X | X | X | X | X | X | X | X | X | X | X |
| HBeAg qualitative | X | | | | | | | | | | | | | |
| HBeAg quantitative | | X | | X | X | X | X | X | X | X | X | X | X | X |
| Anti-HBe qualitative | X | | | | | | | | | | | | | |
| HBV DNA quantification | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HBV genotyping | | X | | | | | | | | | | | | |

| Study Stage | Screening | Treatment Period <sup>a</sup> | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | W1 | | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to D-1 | D1 | D8 ±2 | D29±2 | D57±2 | D85±2 | D113±2 | D141±2 | D169±2 | D197±2 | D225±2 | D253±2 | D281±2 | D309±2 |
| Complement testing <sup>q</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| VIR-3434 PK <sup>s</sup> | | X | X | X | X | X | X | X | | X | | X | | X |
| VIR-3434 immunogenicity <sup>t</sup> | | X | | X | X | X | X | X | X | X | X | X | X | X |
| <b>Exploratory Assessments</b> | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | |

D = day; EOT = end of treatment; W = week

<sup>&</sup>lt;sup>a</sup> On days in which study intervention is administered, assessments performed predose unless otherwise specified.

<sup>&</sup>lt;sup>b</sup> If a participant discontinues treatment or withdraws prematurely from the study prior to the Week 44 visit, EOT assessments should be performed.

<sup>&</sup>lt;sup>c</sup> Prior to study intervention administration on Day 1, participant eligibility will be confirmed.

<sup>&</sup>lt;sup>d</sup> Vital signs (blood pressure, pulse rate, respiratory rate, and temperature) should be measured after the participant has rested comfortably for approximately 10 minutes.

- <sup>e</sup> After signing of the informed consent form (ICF), but prior to initiation of study intervention, AEs/SAEs related to protocol-mandated procedures will be reported. Following initiation of study intervention, all AEs/SAEs, regardless of cause or relationship, will be recorded for the entire duration of the study. Further details can be found in Section 8.7.
- f Does not need to be performed if the participant has had a liver elastography (eg, FibroScan or other sponsor-approved method) in the 6 months prior to screening or liver biopsy in the year prior to screening that confirmed the absence of METAVIR F3 fibrosis or F4 cirrhosis.
- g 12-lead safety ECG will be recorded and should be measured in the supine position after the participant has rested comfortably for approximately 10 minutes. Further details can be found in Section 8.10.
- h Participants will be monitored for ECI, and additional assessments may be performed if indicated. See Section 10.7 and Section 8.7.6 for more information.
- <sup>i</sup> On Day 1, local tolerability should be assessed approximately 1 hour after VIR-3434 administration. At the discretion of the investigator, unscheduled visits are permitted as needed for follow-up of any unresolved local tolerability symptoms. Local tolerability symptoms occurring at other visits should be reported as AEs.
- <sup>j</sup> VIR-3434 will be administered via SC injection. Participants will be monitored for at least 1 hour after VIR-3434 administration.
- <sup>k</sup> TDF will be administered daily orally.

#### CCI

- <sup>m</sup> Screening laboratory tests may be repeated (eg, for values thought to be erroneous) with Sponsor approval.
- <sup>n</sup> WOCBP are required to have pregnancy tests. A blood pregnancy test will be performed at screening, and a urine pregnancy test will be performed at subsequent visits. Negative pregnancy test must be confirmed prior to study intervention administration.
- <sup>o</sup> See Section 8.4 for viral serology parameters.
- <sup>p</sup> Clinical laboratory and urinalysis parameters are described in Section 0.
- <sup>q</sup> Additional samples for urinalysis and complement testing will be collected at any time if fever, rash, or arthralgia are observed in a participant without alternative explanation per the assessment of the investigator, or if immune complex disease is suspected by the investigator based on other signs or symptoms consistent with immune complex disease. Other signs and symptoms consistent with immune complex disease include, but are not limited to, decreased complement, hematuria, proteinuria, and/or decreased renal function. Urinalysis parameters are described in Section 0.
- <sup>r</sup> Drugs of abuse included in the panel are described in Section 0.
- s At all visits during the Treatment Period where PK collection is required, samples will be collected predose only. On Day 8, VIR-3434 will not be dosed, therefore, PK sample can be collected at any time. VIR-3434 PK sample collection includes samples for free and total PK assays, as applicable. Predose samples will be collected within 1 hour prior to dose. Further details can be found in Section 8.8.
- <sup>t</sup> Includes samples for ADA and neutralizing antibodies (NAb), as applicable for VIR-3434. Samples will be collected prior to dosing and at each indicated timepoint thereafter. Additional samples for immunogenicity analysis may be collected if a persistent drug related immunologic event is suspected.
- <sup>u</sup> See Section 8.4 for more information.

#### CCI

#### **CCI**
**Table 9:** Schedule of Activities: Cohort 2b

| Study Stage | Screening | g Treatment Period <sup>a</sup> | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | | v | V1 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to<br>D-1 | D1 | D2 | D8<br>±2 | D29<br>±2 | D57<br>±2 | D85<br>±2 | D113<br>±2 | D141<br>±2 | D169<br>±2 | D197<br>±2 | D225<br>±2 | D253<br>±2 | D281<br>±2 | D309<br>±2 |
| Study procedures | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | Xc | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | |
| Physical examination | X | | | | | | | | | | | | | | X |
| Body weight | | | | | | | | X | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | |
| Vital signs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse event review/record e | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Liver elastography (eg, Fibroscan) f | X | | | | | | | | | | | | | | |
| 12-lead safety ECG <sup>g</sup> | X | | | X | | | | | | | | | | | |
| ECI surveillance h | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| VIR-3434 local tolerability i | | X | | | | | | | | | | | | | |
| Drug Administration | | | | | | | | | | | | | | | |
| VIR-3434 and VIR-2218<br>administration <sup>j</sup> | | X | | | X | X | X | X | X | X | X | X | X | X | X |
| TDF administration (QD) k | | | • | • | • | • | | | X | | • | | | | |

| Study Stage | Screening | ning Treatment Period <sup>a</sup> | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | | v | V1 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to<br>D-1 | | | D8<br>±2 | D29<br>±2 | D57<br>±2 | D85<br>±2 | D113<br>±2 | D141<br>±2 | D169<br>±2 | D197<br>±2 | D225<br>±2 | D253<br>±2 | D281<br>±2 | D309<br>±2 |
| CCI | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | |
| Treatment Diary | | | | | | | | ] | X | | | | | | |
| Laboratory Assessments <sup>m</sup> | | | | | | | | | | | | | | | |
| Pregnancy test <sup>n</sup> | X | X | | X | X | X | X | X | X | X | X | X | X | X | X |
| Screening viral serology o | X | | | | | | | | | | | | | | |
| Liver function tests p | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum chemistry <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation parameters q | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis <sup>pq</sup> | X | X | | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine for drugs of abuse r | X | | | | | | | | | | | | | | |
| HBsAg quantitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Anti-HBs qualitative | X | | | | | | | | | | | | | | |
| Anti-HBs quantitative | | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| HBeAg qualitative | X | | | | | | | | | | | | | | |
| HBeAg quantitative | | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| Anti-HBe qualitative | X | | | | | | | | | | | | | | |
| HBV DNA quantification | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HBV genotyping | | X | | | | | | | | | | | | | |

| Study Stage | Screening | Screening Treatment Period <sup>a</sup> | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | | v | V1 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to<br>D-1 | D1 | D2 | D8<br>±2 | D29<br>±2 | D57<br>±2 | D85<br>±2 | D113<br>±2 | D141<br>±2 | D169<br>±2 | D197<br>±2 | D225<br>±2 | D253<br>±2 | D281<br>±2 | D309<br>±2 |
| Complement testing q | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| VIR-3434 PK predose <sup>s</sup> | | X | | | X | X | X | X | X | | X | | X | | X |
| VIR-3434 PK postdose | | | X <sup>t</sup> | X <sup>u</sup> | | | | | | | | | | | |
| VIR-2218 PK predose <sup>v</sup> | | X | | | | | | | X | | | | | | X |
| VIR-2218 PK postdose | | Xw | Xx | | | | | | Xw | | | | | | X <sup>w</sup> |
| VIR-3434 immunogenicity <sup>y</sup> | | X | | | X | X | X | X | X | X | X | X | X | X | X |
| VIR-2218 immunogenicity <sup>z</sup> | | X | | | X | X | | X | | X | | X | | X | |
| <b>Exploratory Assessments</b> | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | |
| CCI | | | ı | ı | Ī | ı | ı | Ī | ı | ı | | | | | |
| CCI | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | |

| Study Stage | Screening | Treatment Period <sup>a</sup> | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Week | | | W1 | | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44/<br>EOT <sup>b</sup> |
| Visit Day ± Visit Window | D-56 to<br>D-1 | D1 | D2 | D8<br>±2 | D29<br>±2 | D57<br>±2 | D85<br>±2 | D113<br>±2 | D141<br>±2 | D169<br>±2 | D197<br>±2 | D225<br>±2 | D253<br>±2 | D281<br>±2 | D309<br>±2 |
| CCI | | | | | | | | | | | | | | | |

D = day; EOT = end of treatment; W = week

# CCI

<sup>c</sup> Prior to study intervention administration on Day 1, participant eligibility will be confirmed.

### CCI

# **CCI**

- <sup>e</sup> After signing of the informed consent form (ICF), but prior to initiation of study intervention, AEs/SAEs related to protocol-mandated procedures will be reported. Following initiation of study intervention, all AEs/SAEs, regardless of cause or relationship, will be recorded for the entire duration of the study. Further details can be found in Section 8.7
- f Does not need to be performed if the participant has had a liver elastography (eg, FibroScan or other sponsor-approved method) in the 6 months prior to screening or liver biopsy in the year prior to screening that confirmed the absence of Metavir F3 fibrosis or F4 cirrhosis.
- <sup>g</sup> 12-lead safety ECG will be recorded and should be measured in the supine position after the participant has rested comfortably for approximately 10 minutes. Further details can be found in Section 8.10.
- <sup>h</sup> Participants will be monitored for ECI, and additional assessments may be performed if indicated. See Section 10.7 and Section 8.7.6 for more information.
- <sup>i</sup> On Day 1, local tolerability should be assessed approximately 1 hour after VIR-3434 administration. At the discretion of the investigator, unscheduled visits are permitted as needed for follow-up of any unresolved local tolerability symptoms. Local tolerability symptoms occurring at other visits should be reported as AEs.
- <sup>j</sup> VIR-3434 and VIR-2218 will be administered via SC injection. Participants will be monitored for at least 1 hour after VIR-3434 administration.
- <sup>k</sup> TDF will be administered daily orally.
- <sup>1</sup> Patient reported outcomes surveys will be administered as described in Section 8.5.
- <sup>m</sup> Screening laboratory tests may be repeated (eg, for values thought to be erroneous) with Sponsor approval.
- <sup>n</sup> WOCBP are required to have pregnancy tests. A blood pregnancy test will be performed at screening, and a urine pregnancy test will be performed at subsequent visits. Negative pregnancy test must be confirmed prior to study intervention administration.
- <sup>o</sup> See Section 8.4 for viral serology parameters.

<sup>&</sup>lt;sup>a</sup> On days in which study intervention is administered, assessments performed predose unless otherwise specified.

<sup>&</sup>lt;sup>aa</sup> See Section 8.4 for more information.

<sup>&</sup>lt;sup>b</sup> If a participant discontinues treatment or withdraws prematurely from the study prior to the Week 44 visit, EOT assessments should be performed.

- <sup>p</sup> Clinical laboratory and urinalysis parameters are described in Section 0.
- <sup>q</sup> Additional samples for urinalysis and complement testing will be collected at any time if fever, rash, or arthralgia are observed in a participant without alternative explanation per the assessment of the investigator, or if immune complex disease is suspected by the investigator based on other signs or symptoms consistent with immune complex disease. Other signs and symptoms consistent with immune complex disease include, but are not limited to, decreased complement, hematuria, proteinuria, and/or decreased renal function. Urinalysis parameters are described in Section 0.
- <sup>r</sup> Drugs of abuse included in the panel are described in Section 0.
- <sup>s</sup> VIR-3434 PK sample collection includes samples for free and total PK assays, as applicable. Predose samples will be collected within 1 hour prior to dose. Further details can be found in Section 8.8.
- <sup>t</sup> Day 2 VIR-3434 PK postdose sample will be collected between 22 to 28 hours post D1 dose.
- <sup>u</sup> VIR-3434 PK postdose sample can be collected at any time during the D8 visit.
- <sup>v</sup> VIR-2218 PK predose samples will be collected within 1 hour prior to dose. Further details can be found in Section 8.8.
- <sup>w</sup> Day 1, Week 20, and Week 44 VIR-2218 PK postdose samples will be collected between 2 to 6 hours post-dose.
- <sup>x</sup> Day 2 VIR-2218 PK sample will be collected between 22 to 28 hours post D1 dose.
- <sup>y</sup> Includes samples for ADA and neutralizing antibodies (NAb), as applicable for VIR-3434. Samples will be collected prior to dosing and at each indicated timepoint thereafter. Additional samples for immunogenicity analysis may be collected if a persistent drug related immunologic event is suspected.
- <sup>z</sup> Includes samples for ADA of VIR-2218. Samples will be collected prior to dosing and at each indicated timepoint thereafter. Additional samples for immunogenicity analysis may be collected if a persistent drug related immunologic event is suspected.

**Table 10:** Schedule of Activities for Follow-Up Period for all Cohorts

| Study Stage | | | | | | | ] | Follow-U | p Perio | d | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow up Visit | F1 | F2 | F4 | F6 | F8 | F10 | F12 | F16 | F20 | F24 | F28 | F32 | F36 | F40 | F44 | F48/<br>EOFU |
| Visit Day ± Visit<br>Window | D8<br>±2 | D15<br>±2 | D29<br>±7 | D43<br>±7 | D57<br>±7 | D71<br>±7 | D85<br>±7 | D113<br>±7 | D141<br>±7 | D169<br>±7 | D197<br>±7 | D225<br>±7 | D253<br>±7 | D281<br>±7 | D309<br>±7 | D337<br>± 7 |
| Study Procedures | | | | | | | | | | | | | | | | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse event<br>review/record <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead safety ECG <sup>b</sup> | X | | | | | | | | | | | | | | | |
| ECI surveillance <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CCI | | | ı | ı | l | l | l | ı | I | | ı | l | | l | l | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| Laboratory Assessme | ents | | 1 | 1 | | | <u> </u> | 1 | | | 1 | | | | <u> </u> | <u> </u> |
| Pregnancy test <sup>e</sup> | X | | X | | X | | X | | | | | | | | | X |
| Liver function tests <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum chemistry <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation<br>parameters <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis <sup>fg</sup> | X | | X | | X | | X | | | | | | | | | |
| HBsAg quantitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| Study Stage | Follow-Up Period | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow up Visit | F1 | F2 | F4 | F6 | F8 | F10 | F12 | F16 | F20 | F24 | F28 | F32 | F36 | F40 | F44 | F48/<br>EOFU |
| Visit Day ± Visit<br>Window | D8<br>±2 | D15<br>±2 | D29<br>±7 | D43<br>±7 | D57<br>±7 | D71<br>±7 | D85<br>±7 | D113<br>±7 | D141<br>±7 | D169<br>±7 | D197<br>±7 | D225<br>±7 | D253<br>±7 | D281<br>±7 | D309<br>±7 | D337<br>± 7 |
| Anti-HBs quantitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HBeAg quantitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Anti-HBe qualitative | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HBV DNA<br>quantification | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Complement testing <sup>g</sup> | X | | X | | | | | | | | | | | | | |
| VIR-3434 PK <sup>h</sup> | X | | X | | X | | X | X | X | X | | | X | | | X |
| VIR-3434<br>immunogenicity <sup>i</sup> | X | | X | | X | | | X | X | | | | X | | | X |
| VIR-2218<br>immunogenicity <sup>j</sup> | X | | X | | X | | | X | X | | | | X | | | X |
| Exploratory Assessme | ents | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | i | | i | | | i | i | | | i | i | | i | i | | |

| Study Stage | Follow-Up Period | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow up Visit | F1 | F2 | F4 | F6 | F8 | F10 | F12 | F16 | F20 | F24 | F28 | F32 | F36 | F40 | F44 | F48/<br>EOFU |
| Visit Day ± Visit<br>Window | D8<br>±2 | D15<br>±2 | D29<br>±7 | D43<br>±7 | D57<br>±7 | D71<br>±7 | D85<br>±7 | D113<br>±7 | D141<br>±7 | D169<br>±7 | D197<br>±7 | D225<br>±7 | D253<br>±7 | D281<br>±7 | D309<br>±7 | D337<br>± 7 |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |

D = day; EOFU = End of Follow-Up; F = Follow-Up Week

### CCI

- <sup>e</sup> WOCBP are required to have pregnancy tests. A urine pregnancy test will be performed.
- <sup>f</sup> Clinical laboratory and urinalysis parameters are described in Section 0.
- g Additional samples for urinalysis and complement testing will be collected at any time if fever, rash, or arthralgia are observed in a participant without alternative explanation per the assessment of the investigator, or if immune complex disease is suspected by the investigator based on other signs or symptoms consistent with immune complex disease. Other signs and symptoms consistent with immune complex disease include, but are not limited to, decreased complement, hematuria, proteinuria, and/or decreased renal function. Urinalysis parameters are described in Section 0.
- h VIR-3434 PK sample collection includes samples for free and total PK assays, as applicable. Further details can be found in Section 8.8.
- <sup>i</sup> Includes samples for ADA and neutralizing antibodies (NAb), as applicable for VIR-3434. Additional samples for immunogenicity analysis may be collected if a persistent immunologic related event is suspected.
- j Includes samples for ADA of VIR-2218. Additional samples for immunogenicity analysis may be collected if a persistent drug related immunologic event is suspected.
- <sup>k</sup> See Section 8.4 for more information.

| CCI |
|-----|
| CCI |

<sup>&</sup>lt;sup>a</sup> In the Follow-Up Period, all AEs/SAEs, regardless of cause or relationship, will be recorded for the entire duration of the study. Further details can be found in Section 8.7.

<sup>&</sup>lt;sup>b</sup> 12-lead safety ECG will be recorded and should be measured in the supine position after the participant has rested comfortably for approximately 10 minutes. Further details can be found in Section 8.10.

<sup>&</sup>lt;sup>c</sup> Participants will be monitored for ECI, and additional assessments may be performed if indicated. See Section 10.7 for more information.

# 11. REFERENCES

Agarwal K, Yuen M, Wedemeyer, H, et al. Dose-dependent durability of hepatitis B surface antigen reductions following administration of a single dose of VIR-3434, a novel neutralizing vaccinal monoclonal antibody. EASL International Liver Congress, June 22-26, 2022.

Agarwal K, Yuen MF, Wedemeyer H, Arizpe A, et al. Rapid HBsAg Reduction in Chronic Hepatitis B Virus Infection: Preliminary Results From a Phase 1 Study Evaluating a Single Dose of VIR-3434, a Novel Neutralizing, Vaccinal Monoclonal Antibody. Poster. Presented at AASLD: The Liver Meeting (Virtual), November 12-15, 2021.

Ahn SH, Marcellin P, Ma X, Caruntu FA, Tak WY, Elkhashab M, Chuang WL, Tabak F, Mehta R, Petersen J, Guyer W, Jump B, Chan A, Subramanian M, Crans G, Fung S, Buti M, Gaeta GB, Hui AJ, Papatheodoridis G, Flisiak R, Chan HLY. Hepatitis B Surface Antigen Loss with Tenofovir Disoproxil Fumarate Plus Peginterferon Alfa-2a: Week 120 Analysis. Dig Dis Sci. 2018 Dec;63(12):3487-3497. doi: 10.1007/s10620-018-5251-9. Epub 2018 Aug 22. Erratum in: Dig Dis Sci. 2018 Oct 15;: PMID: 30136045; PMCID: PMC6244971.

Bang YJ, Giaccone G, Im SA, Oh DY, Bauer TM, Nordstrom JL, Li H, Chichili GR, Moore PA, Hong S, Stewart SJ, Baughman JE, Lechleider RJ, Burris HA. First-in-human phase 1 study of margetuximab (MGAH22), an Fc-modified chimeric monoclonal antibody, in patients with HER2-positive advanced solid tumors. Ann Oncol. 2017 Apr 1;28(4):855-861. doi: 10.1093/annonc/mdx002. PMID: 28119295; PMCID: PMC6246722.

Bengsch B, Martin B, Thimme R. Restoration of HBV-specific CD8+ T cell function by PD-1 blockade in inactive carrier patients is linked to T cell differentiation. J Hepatol. 2014 Dec;61(6):1212-9. doi: 10.1016/j.jhep.2014.07.005. Epub 2014 Jul 10. PMID: 25016223.

Bertoletti A, Ferrari C. Adaptive immunity in HBV infection. J Hepatol. 2016 Apr;64(1 Suppl):S71-S83. doi: 10.1016/j.jhep.2016.01.026. PMID: 27084039.

Björnsson ES. Hepatotoxicity by Drugs: The Most Common Implicated Agents. Int J Mol Sci2016 Feb 6;17(2):224. doi: 10.3390/ijms17020224. PMID: 26861310; PMCID: PMC4783956.

Burton AR, Pallett LJ, McCoy L, et al. Dysfunctional surface antigen-specific memory B cells accumulate in chronic hepatitis B infection. European Association for the Study of the Liver International Liver Congress 2018. Paris, France.

DiLillo DJ, Ravetch JV. Differential Fc-Receptor Engagement Drives an Anti-tumor Vaccinal Effect. Cell. 2015 May 21;161(5):1035-1045. doi: 10.1016/j.cell.2015.04.016. Epub 2015 May 11. PMID: 25976835; PMCID: PMC4441863.

European Association for the Study of the Liver. Electronic address: easloffice@easloffice.eu; European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID: 28427875.

FDA. Chronic Hepatitis B Virus Infection: Developing Drugs for Treatment. https://www.fda.gov/media/117977/download. Apr 2022.

Galun E, Eren R, Safadi R, Ashour Y, Terrault N, Keeffe EB, Matot E, Mizrachi S, Terkieltaub D, Zohar M, Lubin I, Gopher J, Shouval D, Dagan S. Clinical evaluation (phase I) of a combination of two human monoclonal antibodies to HBV: safety and antiviral properties. Hepatology. 2002 Mar;35(3):673-9. doi: 10.1053/jhep.2002.31867. Erratum in: Hepatology 2002 Apr;35(4):986. PMID: 11870383.

Gane E, Lim YS, Cloutier D, Shen L, et al. Safety and Antiviral Activity of VIR-2218, An X-Targeting RNAi Therapeutic, In Participants With Chronic Hepatitis B Infection: Week 48 Follow-Up Results. Oral Presentation. Presented at the EASL Digital International Liver Conference, June 23-26, 2021.

Gaudinski MR, Coates EE, Houser KV, Chen GL, Yamshchikov G, Saunders JG, Holman LA, Gordon I, Plummer S, Hendel CS, Conan-Cibotti M, Lorenzo MG, Sitar S, Carlton K, Laurencot C, Bailer RT, Narpala S, McDermott AB, Namboodiri AM, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 606 Study Team. Safety and pharmacokinetics of the Fc-modified HIV-1 human monoclonal antibody VRC01LS: A Phase 1 open-label clinical trial in healthy adults. PLoS Med. 2018 Jan 24;15(1):e1002493. doi: 10.1371/journal.pmed.1002493. PMID: 29364886; PMCID: PMC5783347.

Gupta SV, Arizpe A, Fanget M, Dholakiya SL, et al. Preliminary Pharmacokinetics and Safety in Healthy Volunteers of VIR-3434, a Monoclonal Antibody for the Treatment of Chronic Hepatitis B Infection. Poster. Presented at the EASL Digital International Liver Conference, June 23–26, 2021.

Im S-A, Bang Y-J, Oh D-Y, Giaccone G., Bauer T, Nordstrom J, Li H, Moore P, Hong S, Baughman J, Rock E, BurrisH. Long-term responders to single-agent margetuximab, an Fc-modified anti-HER2 monoclonal antibody, in metastatic HER2+ breast cancer patients with prior anti-HER2 therapy. DOI: 10.1158/1538-7445.SABCS18-P6-18-11 Published February 2019.

Invernizzi F, Viganò M, Grossi G, Lampertico P. The prognosis and management of inactive HBV carriers. Liver Int. 2016 Jan;36 Suppl 1:100-4. doi: 10.1111/liv.13006. PMID: 26725905.

Ko SY, Pegu A, Rudicell RS, Yang ZY, Joyce MG, Chen X, Wang K, Bao S, Kraemer TD, Rath T, Zeng M, Schmidt SD, Todd JP, Penzak SR, Saunders KO, Nason MC, Haase AT, Rao SS, Blumberg RS, Mascola JR, Nabel GJ. Enhanced neonatal Fc receptor function improves protection against primate SHIV infection. Nature. 2014 Oct 30;514(7524):642-5. doi: 10.1038/nature13612. Epub 2014 Aug 13. PMID: 25119033; PMCID: PMC4433741.

Lee HW, Park JY, Hong T, et al. A prospective, open-label, dose-escalation, single-center, phase 1 study for GC1102, a recombinant human immunoglobulin for chronic hepatitis B patients. American Association for the Study of Liver Diseases. The Liver Meeting 2018. Abstract 453.

Lim YS, Yuen MF, Cloutier D, Thanawala V, Shen L, Gupta SV, Arizpe A, Cathcart A, Hwang C, Gane E. Longer Treatment Duration of Monthly VIR-2218 Results in Deeper and More Sustained Reductions in Hepatitis B Surface Antigen in Participants with Chronic Hepatitis B Infection. Oral Presentation. Presented at EASL International Liver Conference, June 22-26, 2022.

Maini MK, Gehring AJ. The role of innate immunity in the immunopathology and treatment of HBV infection. J Hepatol. 2016 Apr;64(1 Suppl):S60-S70. doi: 10.1016/j.jhep.2016.01.028. PMID: 27084038.

Marcellin P, Ahn SH, Ma X, Caruntu FA, Tak WY, Elkashab M, Chuang WL, Lim SG, Tabak F, Mehta R, Petersen J, Foster GR, Lou L, Martins EB, Dinh P, Lin L, Corsa A, Charuworn P, Subramanian GM, Reiser H, Reesink HW, Fung S, Strasser SI, Trinh H, Buti M, Gaeta GB, Hui AJ, Papatheodoridis G, Flisiak R, Chan HL; Study 149 Investigators. Combination of Tenofovir Disoproxil Fumarate and Peginterferon α-2a Increases Loss of Hepatitis B Surface Antigen in Patients With Chronic Hepatitis B. Gastroenterology. 2016 Jan;150(1):134-144.e10. doi: 10.1053/j.gastro.2015.09.043. Epub 2015 Oct 8. PMID: 26453773.

Perrillo R, Buti M, Durand F, Charlton M, Gadano A, Cantisani G, et al. Entecavir and hepatitis B immune globulin in patients undergoing liver transplantation for chronic hepatitis B. Liver Transpl. 2013 Aug;19(8):887–95.

Pondé NF, Lambertini M, de Azambuja E. Twenty years of anti-HER2 therapy-associated cardiotoxicity. ESMO Open. 2016 Jul 21;1(4):e000073. doi: 10.1136/esmoopen-2016-000073. PMID: 27843627; PMCID: PMC5070246.

Reed WD, Eddleston AL, Cullens H, Williams R, Zuckerman AJ, Peters DK, Williams DG, Maycock WA. Infusion of hepatitis-B antibody in antigen-positive active chronic hepatitis. Lancet. 1973 Dec 15;2(7842):1347-51. doi: 10.1016/s0140-6736(73)93321-7. PMID: 4128052.

Revill PA, Penicaud C, Brechot C, Zoulim F. Meeting the Challenge of Eliminating Chronic Hepatitis B Infection. Genes (Basel). 2019 Apr 1;10(4):260. doi: 10.3390/genes10040260. PMID: 30939846; PMCID: PMC6523454.

Riccio G, Coppola C, Piscopo G, Capasso I, Maurea C, Esposito E, De Lorenzo C, Maurea N. Trastuzumab and target-therapy side effects: Is still valid to differentiate anthracycline Type I from Type II cardiomyopathies? Hum Vaccin Immunother. 2016 May 3;12(5):1124-31. doi: 10.1080/21645515.2015.1125056. Epub 2016 Feb 2. PMID: 26836985; PMCID: PMC4963071.

Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID: 26563120; PMCID: PMC4722087.

Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. PMID: 29405329; PMCID: PMC5975958.

Trepo C. A brief history of hepatitis milestones. Liver Int. 2014 Feb;34 Suppl 1:29-37. doi: 10.1111/liv.12409. PMID: 24373076.

Tsuge M, Hiraga N, Uchida T, Kan H, Miyaki E, Masaki K, Ono A, Nakahara T, Abe-Chayama H, Zhang Y, Naswa MG, Kawaoka T, Miki D, Imamura M, Kawakami Y, Aikata H, Ochi H, Hayes CN, Chayama K. Antiviral effects of anti-HBs immunoglobulin and vaccine on HBs antigen seroclearance for chronic hepatitis B infection. J Gastroenterol. 2016 Nov;51(11):1073-1080. doi: 10.1007/s00535-016-1189-x. Epub 2016 Mar 4. PMID: 26943168.

Yeo YH, Tseng TC, Hosaka T, Cunningham C, Fung JYY, Ho HJ, Kwak MS, Trinh HN, Ungtrakul T, Yu ML, Kobayashi M, Le AK, Henry L, Li J, Zhang J, Sriprayoon T, Jeong D,

Tanwandee T, Gane E, Cheung RC, Wu CY, Lok AS, Lee HS, Suzuki F, Yuen MF, Kao JH, Yang HI, Nguyen MH. Incidence, Factors, and Patient-Level Data for Spontaneous HBsAg Seroclearance: A Cohort Study of 11,264 Patients. Clin Transl Gastroenterol. 2020 Sep;11(9):e00196. doi: 10.14309/ctg.0000000000000196. PMID: 33094953; PMCID: PMC7494149.

VIREAD® (tenofovir disoproxil fumarate) [US package insert]. Foster City, CA: Gilead Sciences, Inc.; 2019.

Yuen MF, Lim YS, Cloutier D, Thanawala V, et al. Preliminary Results From a Phase 2 Study Evaluating VIR-2218 Alone and in Combination With Pegylated Interferon Alfa-2a in Participants With Chronic Hepatitis B Infection. Oral Presentation. Presented at AASLD: The Liver Meeting (Virtual), November12-15, 2021.

Zalevsky J, Chamberlain AK, Horton HM, Karki S, Leung IW, Sproule TJ, Lazar GA, Roopenian DC, Desjarlais JR. Enhanced antibody half-life improves in vivo activity. Nat Biotechnol. 2010 Feb;28(2):157-9. doi: 10.1038/nbt.1601. Epub 2010 Jan 17. PMID: 20081867; PMCID: PMC2855492.

Zoulim F, Durantel D. Antiviral therapies and prospects for a cure of chronic hepatitis B. Cold Spring Harb Perspect Med. 2015 Apr 1;5(4):a021501. doi: 10.1101/cshperspect.a021501. PMID: 25833942; PMCID: PMC4382723.

| · · |
|-----|

PPD